CLINICAL TRIAL: NCT03807440
Title: CORDIALLY® - CEE: Characteristics of Patients With Type 2 Diabetes Treated With Modern Antidiabetic Drugs. A Real World Data Collection of Patient Baseline Characteristics, Treatment Patterns and Comorbidities in Central Eastern European (CEE) Countries
Brief Title: DIA_CENTRAL:T2D Treatment Pattern in Central Europe
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1245-0187
Record Dates: First submitted 2019-01-15; First posted 2019-01-17 (Actual); Results first posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; Sodium-Glucose Transporter 2 Inhibitors; Dipeptidyl-Peptidase IV Inhibitors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with Diabetes Mellitus, Type 2
  Interventions: Drug: Empagliflozin; Drug: Sodium Glucose Transporter 2 inhibitor; Drug: Dipeptidyl-peptidase 4 inhibitor; Drug: Glucagon-like peptide 1 agonist

INTERVENTIONS:
Drug: Empagliflozin — Empagliflozin
  Other Names: Jardiance® Synjardy® Trajenta® Jentadueto®
Drug: Sodium Glucose Transporter 2 inhibitor — Sodium Glucose Transporter 2 inhibitor
  Other Names: Jardiance® Synjardy® Trajenta® Jentadueto®
Drug: Dipeptidyl-peptidase 4 inhibitor — Dipeptidyl-peptidase 4 inhibitor
  Other Names: Jardiance® Synjardy® Trajenta® Jentadueto®
Drug: Glucagon-like peptide 1 agonist — Glucagon-like peptide 1 agonist
  Other Names: Jardiance® Synjardy® Trajenta® Jentadueto®

SUMMARY:
This is a non-interventional study using existing data including medical chart review.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to participation
2. Female and male patients age ≥ 18 years
3. Patients with T2D diagnosis
4. Patients who have been newly initiated (first ever use) with empagliflozin or other Sodium Glucose Transporter 2 inhibitor (SGLT2i), Dipeptidyl-peptidase 4 inhibitor (DPP4i) or Glucagon-like peptide 1 agonist (GLP1a) between September 2018 and December 2018 (study index date 1)
5. Patients have been naïve to treatment with empagliflozin or other Sodium Glucose Transporter 2 inhibitor (SGLT2i), Dipeptidyl-peptidase 4 inhibitor (DPP4i) or Glucagon-like peptide 1 agonist (GLP1a) at study index date 1

Exclusion Criteria:

1. Patients age < 18 years
2. Patients with diagnosis of other types of diabetes than T2D
3. Patients who do not provide written consent to the terms of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (18 years of age or older) with Type 2 Diabetes diagnosis, naïve to treatment with empagliflozin or other Sodium Glucose Transporter 2 inhibitor (SGLT2i), DPP4i (Dipeptidyl-peptidase 4 inhibitor) or GLP1a (Glucagon-like peptide 1 agonist) at index date were chosen.
Sampling Method: Non-Probability Sample
Enrollment: 4083 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Medvedchikov, +43180105-7896, Study Chair — Alexey.Medvedchikov@Boehringer-Ingelheim.com
Locations (177):
- Bulgaria (15):
  - MHAT "Julia Verevska-Byala" EOOD, Center Nr.: 35903, Byala
  - MC "Diamedical 2013" OOD, Center Nr.: 35902, Dimitrovgrad
  - MBAL- Dobrich AD, Center Nr.: 35916, Dobrich
  - Dr. T. K. Bacheva - ASMP-IP-E EOOD, Center Nr.: 35904, Dupnitsa
  - MHAT "Medline Clinic", Center Nr.: 35911, Plovdiv
  - MC Kuchuk Parij OOD, Center Nr.: 35906, Plovdiv
  - MC Saint Elisaveta-Rakovski EOOD, Center Nr.: 35909, Rakovski
  - "Medical Center-Razgrad"OOD, Center Nr.: 35910, Razgrad
  - DCC 1 - Russe EOOD, Center Nr.: 35905, Rousse
  - MBAL "Hadzhi Dimitar" OOD, Center Nr.: 35915, Sliven
  - MC Polimed AD, Center Nr.: 35907, Sofia
  - MC Gina - LZ SIMP EOOD, Center Nr.: 35918, Sofia
  - MC "Vitaclinic" EOOD, Center Nr.: 35901, Sofia
  - MC Kalimat EOOD, Center Nr.: 35914, Sofia
  - Acibadem City Clinic Medical Center Varna EOOD, Center Nr.: 35908, Varna
- Czechia (58):
  - Michal Brada, Center Nr.: 42001, Beclav
  - Dr. Kovaová, Center Nr.: 42069, Beroun
  - Practice Dr. Alice Sýkorová, Center Nr.: 42057, Bílina
  - MUDr. Alica Vesela, Center Nr.: 42030, Broumov
  - EUC Klinika eské Budjovice, Center Nr.: 42052, Eské Budjovice
  - Lékaský dm Géko, Center Nr.: 42059, Eské Budjovice
  - Barbara Buzová, Center Nr.: 42003, Havíov
  - Zaviatiová, Petra, Center Nr.: 42004, Havíov
  - Radana Syslová, Center Nr.: 42035, Hlušovice
  - Pavel Kasík, Center Nr.: 42046, Hoovice
  - Practice Dr. Petr Maule, Center Nr.: 42054, Humpolec
  - Mediab Jihlava s.r.o., Center Nr.: 42066, Jihlava
  - Practice MUDr. Gita Markofová, Center Nr.: 42053, Karlovy Vary
  - Dr. Konená, Center Nr.: 42036, Karviná - Staré Msto
  - Practice Zdzislaw Wranka, Center Nr.: 42072, Karviná-Hranice
  - Pavel Tománek, Center Nr.: 42028, Kopivnice
  - DIABET HELP s.r.o., Center Nr.: 42058, Kralupy nad Vltavou
  - MUDr.Tomáš Edelsberger, Center Nr.: 42007, Krnov
  - Jitka Hasalová, Center Nr.: 42010, Kromiz
  - árka Drinková, Center Nr.: 42038, Lede Nad Sázavou
  - Martina Košková, Center Nr.: 42047, Mladá Boleslav
  - Dobromila Vykoupilová, Center Nr.: 42033, Nmice Nad Hanou
  - Karel Churavý, Center Nr.: 42005, Nový Jiín
  - árka Kubánková, Center Nr.: 42048, Nymburk
  - Agentura Science Pro spol. s.r.o., Center Nr.: 42002, Olomouc
  - Anna Rancová, Center Nr.: 42025, Olomouc
  - Josef íný, Center Nr.: 42026, Opava
  - MUDr.Tomáš Hrdina, Center Nr.: 42015, Opono
  - Dr. Šeptáková, Center Nr.: 42074, Ostrava
  - Practice Dr. René Turínek, Center Nr.: 42034, Ostrava
  - MUDr. Eva Raická, Center Nr.: 42024, Ostrava
  - Jitka Homolová, Center Nr.: 42012, Ostrava
  - Radka Nágelová, Center Nr.: 42020, Ostrava Poruba
  - AIDIN VK s.r.o., Center Nr.: 42017, Perov
  - MUDr. Vra Prýmková, Center Nr.: 42070, Píbram
  - Zdenk Jankovec, Center Nr.: 42044, Plze
  - Diabetologická a interní ambulance, Center Nr.: 42064, Podbrady
  - MUDr. Jana Houdová, Center Nr.: 42068, Prague
  - Practice Dr. Milena Peterková, Center Nr.: 42063, Prague
  - MUDr.Michala Pelikánová s.r.o., Center Nr.: 42055, Prague
  - Markéta Hovorková, Center Nr.: 42042, Prague
  - Jakub Hron, Center Nr.: 42043, Prague
  - Milan Fleka, Center Nr.: 42041, Prague
  - Jií Jón, Center Nr.: 42045, Prague
  - Practice Dr. Lucie Kufová, Center Nr.: 42062, Prague
  - Practice Dr. Ida Reissová, Center Nr.: 42056, Prague
  - Barbora Diepoltová, Center Nr.: 42037, Prague
  - Practice Dr. Petronela Janeková, Center Nr.: 42065, Rumburk
  - Practice Dr. Miroslav Lindovský, Center Nr.: 42051, Sokolov
  - Dana Fialkoviová, Center Nr.: 42040, Strakonice
  - Marek Frydrych, Center Nr.: 42008, Tebí
  - Marek Frydrych, Center Nr.: 42077, Tebí
  - Diabetologická ambulance s.r.o., Center Nr.: 42076, Uherské Hradišt
  - Dr. Hrmová, Center Nr.: 42073, Vlašim
  - Lubomír Kudlej, Center Nr.: 42050, Vrchlabí
  - AdiaMed s.r.o., Center Nr.: 42009, Vsetín
  - EUC Klinika Zlín a.s., Center Nr.: 42075, Zlín
  - Robin Urbánek, Center Nr.: 42029, Zlín
- Hungary (10):
  - Bajcsy-Zsilinszky Kórház és Rendelintézet, Center Nr.: 36019, Budapest
  - Jahn Ferenc Dél-pesti Kórház és Rendelintézet, Center Nr.: 36014, Budapest
  - Debreceni Egyetem Klinikai Központ, Kardiológiai Klinika, Center Nr.: 36006, Debrecen
  - Kátai Gábor Kórház, Diabetológia Szakrendelés, Center Nr.: 36007, Karcag
  - Practice Dr. Lelkesi Anita, Center Nr.: 36013, Mátészalka
  - Nagyatádi Kórház, Center Nr.: 36021, Nagyatád
  - Nyírségi Diabetes Centrum, Center Nr.: 36024, Nyíregyháza
  - Dr. Wagner Zoltán, Center Nr.: 36020, Pécs
  - Siófoki Kórház Rendelintézet, Center Nr.: 36004, Siófok
  - Soproni Gyógyközpont, Center Nr.: 36018, Sopron
- Poland (28):
  - Gabinet Diabetologiczno- Internistyczny Katarzyna Wasilewska, Center Nr.: 48011, Biaystok
  - NZOZ DIAMED Sp. z o.o., Center Nr.: 48061, Czechowice-Dziedzice
  - Prywatny Gabinet Lekarski dr n. med. Joanna Sawer-Szewczyk, Center Nr.: 48055, Czyca
  - Zespó Opieki Zdrowotnej w czycy, Center Nr.: 48054, Czyca
  - NZOZ Sal Med, Center Nr.: 48047, Dzieroniów
  - Poradnia Diabetologiczna, Center Nr.: 48028, Gorlice
  - Indywidualna Specjalistyczna Praktyka Lekarska Piotr Piskozub Specjalista Diabetolog, Center Nr.: 48042, Jelenia Góra
  - NZOZ Poradnia Diabetologiczna, Center Nr.: 48038, Konin
  - Zakad Opieki Medycznej Sanatio; Sp. Z. o.o., Center Nr.: 48030, Krakow
  - Prywatny Gabinet Lekarski Tomasz Wierzykowski, Center Nr.: 48053, Kutno
  - Indywidualna Specjalistyczna Praktyka Lekarska Magorzata Poskoska-Lemaska, Center Nr.: 48035, Kwidzyn
  - Indywidualna Specjalistyczna Praktyka Lekarska Barbara Soróbka, Center Nr.: 48001, Legnica
  - Poradnia Cukrzycowa SP ZOZ w Lesku, Center Nr.: 48024, Lesko
  - Lumed Sp. z o.o., Center Nr.: 48032, Lubaczów
  - DIABETA-CARE Sp.z o.o., Center Nr.: 48008, Lubin
  - Poradnia Diabetologiczna Dr. mudziska, Center Nr.: 48013, Nako Nad Noteci
  - Alfa Specjalistyczne Gabinety Lekarskie Ewa Moroz, Center Nr.: 48007, Nowy Scz
  - Poradnia Diabetologiczna Dr. Adamczyk-Gajda, Center Nr.: 48031, Olenica
  - MED-ART Sp. z o.o., Center Nr.: 48052, Orzesze
  - Indywidualna Specjalistyczna Praktyka Lekarska Wiesawa Fischer, Center Nr.: 48020, Ostrów Wielkopolski
  - Prywatny Gabinet Lekarski azuka, Center Nr.: 48026, Parczew
  - Powiatowy Szpital Specjalistyczny w Stalowej Woli, Center Nr.: 48056, Stalowa Wola
  - Prywatny Gabinet Lekarski dr n. med. Piotr Gryglas, Center Nr.: 48059, Warsaw
  - Poradnia Diabetologiczna Szpitala Powiatowego w Wicborku, Center Nr.: 48003, Wicbork
  - Orodek Praktyka Lekarska Konrad Strzelczyk, Center Nr.: 48012, Woomin
  - Poradnia Diabetologiczna SPZZOZ w Wyszkowie, Center Nr.: 48067, Wyszków
  - Wojewódzka Poradnia dla Chorych na Cukrzyc, Center Nr.: 48025, Zabrze
  - Cardiomed, Center Nr.: 48019, Zielona Góra
- Russia (66):
  - Anturium, Center Nr.: 70036, Barnaul
  - Central city hospital, Center Nr.: 70073, Bataysk
  - Chelyabinsk regional clinical hospital, Center Nr.: 70069, Chelyabinsk
  - Russian Medical Academy of Continuing Professional Education, Center Nr.: 70058, Irkutsk
  - The First Republican Clinical Hospital of the Ministry of Health of the Udmurt Republic, Center Nr.: 70037, Izhevsk
  - Central City Hospital No. 18, Center Nr.: 70051, Kazan'
  - Kemerovo regional clinical hospital named S.V. Belyaev, Center Nr.: 70008, Kemerovo
  - City Polyclinic No. 16, Center Nr.: 70067, Khabarovsk
  - Kirov Clinical Hospital No. 7 named after V.I. Yurlova, Center Nr.: 70089, Kirov
  - Krai clinical hospital Nr. 1 named after prof. S.V. Ochapovskogo, Center Nr.: 70049, Krasnodar
  - Lipetsk Regional Hospital, Center Nr.: 70046, Lipetsk
  - SBIH Center for Speech Pathology and Neurorehabilitation MDH, Center Nr.: 70080, Moscow
  - Clinical Hospital No. 85 of trhe Federal Biomedical Agency, Center Nr.: 70042, Moscow
  - National Medical Research Center for Endocrinology, Center Nr.: 70025, Moscow
  - City Polyclinic No. 22 of the Department of Healthcare of the Moscow City, Center Nr.: 70043, Moscow
  - City Polyclinic No. 22 of the Department of Healthcare of the Moscow City, Center Nr.: 70045, Moscow
  - Endocrinology Dispensary of the Moscow City Healthcare Department, Center Nr.: 70032, Moscow
  - Endocrinology Dispensary of the Moscow City Healthcare Department, Center Nr.: 70041, Moscow
  - Endocrinology Dispensary of the Moscow City Healthcare Department, Center Nr.: 70081, Moscow
  - Endocrinology Dispensary of the Moscow City Healthcare Department, Center Nr.: 70084, Moscow
  - Vessel Clinic, Center Nr.: 70011, Moscow
  - City Polyclinic No 107 of the Moscow City Healthcare Department, Center Nr.: 70082, Moscow
  - City Clinical Hospital named after V.V. Veresaeva of the Moscow Department of Health, Center Nr.: 70003, Moscow
  - City Polyclinic No. 1, Center Nr.: 70074, Nal'chik
  - City clinical hospital #12 of Sormovskiy district of Nizhniy Novgorod, Center Nr.: 70018, Nizhny Novgorod
  - Privolzhsky Research Medical University, Center Nr.: 70085, Nizhny Novgorod
  - Novokuznetsk City Clinical Hospital No. 1, Center Nr.: 70050, Novokuznetsk
  - AVICENNA, Center Nr.: 70065, Novosibirsk
  - City Clinical Polyclinic #16, Center Nr.: 70056, Novosibirsk
  - Novosibirsk State Medical University, Center Nr.: 70059, Novosibirsk
  - AVICENNA, Center Nr.: 70064, Novosibirsk
  - Penza regional clinical hospital named after N.N. Burdenko, Center Nr.: 70095, Penza
  - Private Clinic Salon Roden, Center Nr.: 70086, Perm
  - City clinical hospital 5, Center Nr.: 70057, Perm
  - City clinical hospital 5, Center Nr.: 70070, Perm
  - City polyclinic #16 of the City Rostov-on-Don, Center Nr.: 70027, Rostov-on-Don
  - North-West State Medical University named after II. Mechnikov, Center Nr.: 70053, Saint Petersbug
  - North-West State Medical University named after II. Mechnikov, Center Nr.: 70077, Saint Petersbug
  - First Saint-Petersburg state medical university named after acad. I.P.Pavlov, Center Nr.: 70024, Saint Petersburg
  - First Saint-Petersburg state medical university named after acad. I.P.Pavlov, Center Nr.: 70087, Saint Petersburg
  - Medilux-TM, Center Nr.: 70005, Saint Petersburg
  - V.A. Almazov National Medical Research Center, Center Nr.: 70071, Saint Petersburg
  - AntMed, Center Nr.: 70034, Saint Petersburg
  - Dr. Tsiberkin, Center Nr.: 70048, Saint Petersburg
  - City Pokrovskaya Hospital, Center Nr.: 70022, Saint Petersburg
  - Zabotlivyi Doktor, Center Nr.: 70016, Saint Petersburg
  - Samara city polyclinic Nr. 9 of Oktyabrskiy district, Center Nr.: 70028, Samara
  - Samara city consulting and diagnostic polyclinic nr. 14, Center Nr.: 70029, Samara
  - Clinical Hospital of the Saratov city, Center Nr.: 70090, Saratov
  - LLC clinic "Family Doctor", Center Nr.: 70093, Saratov
  - Multifunctional Medical Clinic "Sova", Center Nr.: 70030, Saratov
  - Regional Endocrinological Dispensary, Center Nr.: 70078, Stavropol
  - Tyumen State Medical University, Center Nr.: 70066, Tyumen
  - City clinical hospital, Center Nr.: 70019, Ufa
  - City Polyclinic No.2, Center Nr.: 70062, Ulan-Ude
  - Limited Liability Company "CENTER", Center Nr.: 70060, Vladivostok
  - Regional Clinical Hospital No. 2, Center Nr.: 70092, Vladivostok
  - Regional Clinical Hospital No. 2, Center Nr.: 70068, Vladivostok
  - Volgograd Regional Clinical Hospital No. 3, Center Nr.: 70076, Volgograd
  - Clinical Polyclinic No.28, Center Nr.: 70040, Volgograd
  - Voronezh City Clinical Hospital #11, Center Nr.: 70035, Voronezh
  - State budgetary institution "City polyclinic Nr. 4", Center Nr.: 70017, Voronezh
  - State budgetary institution "City polyclinic Nr. 4", Center Nr.: 70033, Voronezh
  - State budgetary institution "City polyclinic Nr. 4", Center Nr.: 70055, Voronezh
  - Limited Liability Company "Uralsky Medical Center", Center Nr.: 70063, Yekaterinburg
  - Scientific and Practical Center of Specialized Types of Medical Care "Uralskij Institute of Cardiology", Center Nr.: 70079, Yekaterinburg

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Prazny M, Suplotova L, Gumprecht J, Kamenov Z, Fulop T, Medvedchikov A, Rosenzweig D, Aleksandric M. Real-world characteristics, modern antidiabetic treatment patterns, and comorbidities of patients with type 2 diabetes in central and Eastern Europe: retrospective cross-sectional and longitudinal evaluations in the CORDIALLY(R) study. Cardiovasc Diabetol. 2022 Oct 8;21(1):203. doi: 10.1186/s12933-022-01631-4. PMID 36209118
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a non-interventional, multi-country, multi-site study using existing data from medical records to evaluate treatment pattern of Type 2 Diabetes (T2D) patients under routine conditions. It was conducted in medical practices in Central Eastern Europe (CEE) countries (Bulgaria, Czech Republic, Hungary, Poland, Russian Federation). Healthcare professionals (HCPs) of different specialties involved in treatment of T2D patients participated in this study. In this study .
Pre-assignment Details: Only subjects that met all inclusion and none of the exclusion criteria were included.
  4083 patients were screened, thereof 28 could not be included in the prescribed patient set (PPS).
Groups:
- T2D Patients From Central Eastern Europe: Patients with type 2 diabetes (T2D) from Central Eastern Europe (CEE) (Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who were newly initiated (first ever use) on empagliflozin or other sodium dependent glucose transporter inhibitor (SGLT2i), dipeptidyl peptidase 4 inhibitor (DPP4i) or glucagon-like peptide-1 receptor agonist (GLP-1 RA) between September 2018 and December 2018 (study index date 1).
Period: Overall Study
Arm/Group | T2D Patients From Central Eastern Europe
Started (Patients included in the prescribed patient set (PPS)) | 4055 (Study index date 1)
Completed (Patients included in the full analysis set (FAS)) | 3618 (study index date 2)
Not Completed | 437
Not completed — No documentation of index date 2 | 320
Not completed — No informed consent for index date 2 | 117

BASELINE CHARACTERISTICS:
Population: Prescribed patient set (PPS): All patients fulfilling inclusion and exclusion criteria who have received a first prescription of a respective Type 2 Diabetes (T2D) medication and whose documentation was electronically signed by the physician.
Arm/Group | T2D Patients From Central Eastern Europe
Number analyzed (Participants) | 4055
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age for each patient was calculated by subtracting the year of birth from the year of registration (i.e. Year of registration - Year of birth). Year of registration was defined as the year the patients where initiated on T2D medication.
  Years | 63.1 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1993
  Male | 2062
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 27
  White | 4028
  More than one race | 0
  Unknown or Not Reported | 0
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 169.2 (9.5)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 94.4 (18.8)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram/meter^2 (kg/m^2)] | 32.9 (5.8)
Socioeconomic factor: Employment status [Count of Participants; unit: Participants] — Number of patients in each category of the employment status is reported. The categories of employment status are:
  * Employed;
  * Not employed;
  * Unknown;
  Participants
    Employed | 1930
    Not employed | 1889
    Unknown | 236
Socioeconomic factor: Family status [Count of Participants; unit: Participants] — Number of patients in each category of family status is reported.
  The reported categories of family status are:
  Single; Married; Divorced; Widowed; Unknown;
  Participants
    Single | 278
    Married | 2670
    Divorced | 211
    Widowed | 340
    Unknown | 556
Socioeconomic factor: Insurance status [Count of Participants; unit: Participants] — Number of patients in each category of insurance status is reported.
  The categories of insurance status are:
  * Not insured;
  * Statutory insured;
  * Privately insured;
  * Unknown;
  Participants
    Not insured | 77
    Statutory insured | 3655
    Privately insured | 153
    Unknown | 170
Risk factor for CVD and CKD: Body Mass Index (BMI) categorical [Count of Participants; unit: Participants] — Risk factors for cardiovascular disease (CVD) and chronic kidney disease (CKD): Body Mass Index (BMI) categorical.
  Number of patients in each category of BMI is reported. The reported categories of BMI are:
  * Being obese (BMI ≥30);
  * Being overweight (BMI ≥25 to <30);
  * Being normal (BMI ≥18.5 to ≤24.9);
  * Being underweight <18.5;
  Participants
    Being obese | 2755
    Being overweight | 1086
    Being normal | 212
    Being underweight | 2
Risk factor for CVD and CKD: Hypertension [Count of Participants; unit: Participants] — Risk factor for cardiovascular disease (CVD) and chronic kidney disease (CKD): Hypertension.
  Number of patients with hypertension is reported. Hypertension was defined as systolic blood pressure ≥140 millimetre of mercury (mmHg) and / or diastolic blood pressure ≥90 mmHg.
  Participants
    Yes | 3432
    No | 589
    Unknown | 34
Risk factor for CVD and CKD: Tobacco smoking [Count of Participants; unit: Participants] — Risk factor for cardiovascular disease (CVD) and chronic kidney disease (CKD): Tobacco smoking.
  Number of participants in each category of tobacco smoking is reported.
  The reported categories of tobacco smoking are:
  * Current smoker;
  * Ex-smoker;
  * Never smoker;
  * Unknown;
  Participants
    Current smoker | 664
    Ex-smoker | 933
    Never smoker | 2123
    Unknown | 335
Risk factor for CVD and CKD: Being physically inactive [Count of Participants; unit: Participants] — Risk factor for cardiovascular disease (CVD) and chronic kidney disease (CKD): Being physically inactive. Number of participants in each category of being physically inactive is reported.
  Being physically inactive was defined as less than 2.5 hours of moderate-intensity aerobic exercise or less than 75 minutes of vigorous aerobic exercise per week.
  Participants
    Yes | 2048
    No | 1736
    Unknown | 271
Family history of early heart and kidney disease [Count of Participants; unit: Participants] — Number of patients in each category of family history of early heart disease and family history early kidney disease is reported.
  Participants
    Family history of early heart disease: Yes | 1132
    Family history of early heart disease: No | 1945
    Family history of early heart disease: Unknown | 978
    Family history of early kidney disease: Yes | 266
    Family history of early kidney disease: No | 2609
    Family history of early kidney disease: Unknown | 1180
10 Years Risk for fatal CVD according to the applying SCORE Risk Chart [Mean (Standard Deviation); unit: scale on a score] — 10 Years Risk for fatal cardiovascular disease (CVD) according to the applying Systematic COronary Risk Evaluation (SCORE) Risk Chart (European Society of Cardiology) taking into account patient´s age, gender, systolic blood pressure, smoking status, and total cholesterol value at index date 1.
  SCORE Risk Chart takes values from from 0% to 100%. SCORE Risk Chart values from 5% and upwards indicate a high 10-year risk for a fatal cardiovascular event. Population: Prescribed patient set (PPS): All patients fulfilling inclusion and exclusion criteria who have received a first prescription of a respective Type 2 diabetes (T2D) medication and whose documentation was electronically signed by the physician. Only participants with non-missing results are reported.
  scale on a score
    number analyzed (Participants) | 2613
    (all) | 6.4 (5.5)
Time since diagnosis of type 2 diabetes (T2D) [Mean (Standard Deviation); unit: Years] — Time since diagnosis of type 2 diabetes (T2D) is reported. Time since diagnosis of T2D (years) was calculated by subtracting the year of T2D diagnosis from the year of registration. Year of registration was defined as the year patients where initiated on T2D medication.
  Years | 9.9 (6.9)
Clinical parameter relevant for T2D: HbA1c [Mean (Standard Deviation); unit: millimol/mol] — Clinical parameter relevant for Type 2 Diabetes (T2D): Concentration of glycosylated hemoglobin (HbA1c) Population: Prescribed patient set (PPS): All patients fulfilling inclusion and exclusion criteria who have received a first prescription of a respective T2D medication and whose documentation was electronically signed by the physician. Only participants with non-missing results are reported.
  millimol/mol
    number analyzed (Participants) | 3720
    (all) | 66.8 (14.9)
Clinical parameter relevant for T2D: Glycosylated haemoglobin (HbA1c %) [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] — Clinical parameter relevant for Type 2 Diabetes (T2D): Percentage of glycosylated hemoglobin (HbA1c [%]). Population: Prescribed patient set (PPS): All patients fulfilling inclusion and exclusion criteria who have received a first prescription of a respective T2D medication and whose documentation was electronically signed by the physician. Only participants with non-missing results are reported.
  percentage of glycosylated hemoglobin
    number analyzed (Participants) | 3720
    (all) | 8.3 (1.4)
Clinical parameter relevant for T2D: Glycosylated hemoglobin (HbA1c [%])-categorical [Count of Participants; unit: Participants] — Clinical parameter relevant for Type 2 Diabetes (T2D): Number of patients in each category of glycosylated hemoglobin (HbA1c [%]). The reported categories of HbA1c [%] are:
  * <8.5%;
  * ≥8.5%;
  * Missing;
  Participants
    <8.5% | 2477
    ≥8.5% | 1243
    Missing | 335
Prescribed T2D medication [Count of Participants; unit: Participants] — Number of patients in each category of Type 2 Diabetes medication. The reported categories of Type 2 Diabetes medication are the following:
  * Empagliflozin;
  * Sodium dependent glucose transporter inhibitor (Other SGLT2i);
  * Dipeptidyl peptidase 4 inhibitor (DPP4i);
  * Glucagon-like peptide-1 receptor agonist (GLP-1 RA);
  Participants
    Empagliflozin | 1966
    Other SGLT2i | 584
    DPP4i | 1144
    GLP-1 RA | 361
Prescribed T2D medication [Count of Participants; unit: Participants] — Number of patients for each type of Type 2 Diabetes (T2D) medication.
  Participants
    SGLT2i: Canagliflozin | 156
    SGLT2i: Dapagliflozin | 425
    SGLT2i: Empagliflozin | 1966
    SGLT2i: Ertugliflozin | 3
    DPP4i: Alogliptin | 94
    DPP4i: Linagliptin | 457
    DPP4i: Sitagliptin | 328
    DPP4i: Saxagliptin | 20
    DPP4i: Vildagliptin | 245
    GLP-1 RA: Dulaglutide | 129
    GLP-1 RA: Exenatide | 16
    GLP-1 RA: Liraglutide | 165
    GLP-1 RA: Semaglutide | 2
    GLP-1 RA: Lixisenatide | 49

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients in Each Category of First Prescription of a Respective Modern Type 2 Diabetes (T2D) Medication According to Prescribing Specialist
Description: Number of patients in each category of prescription of a respective modern Type 2 Diabetes (T2D) medication according to prescribing specialist is reported.
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: Prescribed patient set (PPS): All patients fulfilling inclusion and exclusion criteria who have received a first prescription of a respective T2D medication and whose documentation was electronically signed by the physician.
Measure: Count of Participants; unit: Participants
Groups:
- Patients Initiated on T2D Medication by Endocrinologist: Patients with type 2 diabetes (T2D) from Central Eastern Europe (CEE) (Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who were newly initiated (first ever use) on empagliflozin or other sodium dependent glucose transporter inhibitor (SGLT2i), dipeptidyl peptidase 4 inhibitor (DPP4i) or glucagon-like peptide-1 receptor agonist (GLP-1 RA) by endocrinologist between September 2018 and December 2018 (study index date 1).
- Patients Initiated on T2D Medication by Diabetologist: Patients with type 2 diabetes (T2D) from Central Eastern Europe (CEE) (Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who were newly initiated (first ever use) on empagliflozin or other sodium dependent glucose transporter inhibitor (SGLT2i), dipeptidyl peptidase 4 inhibitor (DPP4i) or glucagon-like peptide-1 receptor agonist (GLP-1 RA) by diabetologist between September 2018 and December 2018 (study index date 1).
- Patients Initiated on T2D Medication by Cardiologist: Patients with type 2 diabetes (T2D) from Central Eastern Europe (CEE) (Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who were newly initiated (first ever use) on empagliflozin or other sodium dependent glucose transporter inhibitor (SGLT2i), dipeptidyl peptidase 4 inhibitor (DPP4i) or glucagon-like peptide-1 receptor agonist (GLP-1 RA) by cardiologist between September 2018 and December 2018 (study index date 1).
Arm/Group | Patients Initiated on T2D Medication by Endocrinologist | Patients Initiated on T2D Medication by Diabetologist | Patients Initiated on T2D Medication by Cardiologist
Number analyzed (Participants) | 1652 | 2301 | 102
Participants
  Empagliflozin | 815 | 1073 | 78
  Other SGLT2i | 244 | 333 | 7
  DPP4i | 504 | 624 | 16
  GLP-1 RA | 89 | 271 | 1

2. Primary Outcome: Number of Patients Initiated on a Modern Type 2 Diabetes (T2D) Medication Who Also Received Concomitant T2D Medications at Study Index Date 1 According to Prescribing Specialist
Description: Number of patients initiated on a modern type 2 diabetes (T2D) medication who also received concomitant T2D medications at study index date 1 according to prescribing specialist is reported.
  The concomitant T2D medications reported are:
  * Metformin
  * Sulfonylurea
  * Acarbose
  * Pioglitazone
  * Insulin
  * Others
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on T2D Medication by Endocrinologist | Patients Initiated on T2D Medication by Diabetologist | Patients Initiated on T2D Medication by Cardiologist
Number analyzed (Participants) | 1652 | 2301 | 102
Participants
  Metformin | 1349 | 1794 | 81
  Sulfonylurea | 626 | 513 | 17
  Acarbose | 3 | 49 | 3
  Pioglitazone | 3 | 91 | 0
  Insulin | 342 | 658 | 17
  Others | 59 | 91 | 7

3. Primary Outcome: Number of Patients Initiated on a Modern Type 2 Diabetes (T2D) Medication Who Also Received Concomitant Cardiovascular Disease (CVD) and/or Chronic Kidney Disease (CKD) Medication at Study Index Date 1 According to Prescribing Specialist
Description: Number of patients initiated on a modern type 2 diabetes (T2D) medication who also received concomitant cardiovascular disease (CVD) and/or chronic kidney disease (CKD) medication at study index date 1 according to prescribing specialist is reported.
  The reported concomitant CVD and/or chronic CKD medications are:
  * Antihypertensive angiotensin-converting-enzyme inhibitors (ACEi) or angiotensin II receptor blockers (ARBs)
  * Statins
  * Low dose aspirin
  * Beta blockers
  * Diuretics
  * Others
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on T2D Medication by Endocrinologist | Patients Initiated on T2D Medication by Diabetologist | Patients Initiated on T2D Medication by Cardiologist
Number analyzed (Participants) | 1652 | 2301 | 102
Participants
  Antihypertensive ACEi or ARBs | 1256 | 1536 | 87
  Statins | 983 | 1327 | 82
  Low dose aspirin | 555 | 622 | 64
  Beta blockers | 580 | 922 | 73
  Diuretics | 471 | 732 | 44
  Others | 160 | 455 | 29

4. Primary Outcome: Baseline Characteristic: Age According to Type 2 Diabetes (T2D) Medication for the Patients Who Were Initiated on T2D Medication by Endocrinologist
Description: Baseline characteristic: Age according to type 2 diabetes (T2D) medication for the patients who were initiated on T2D medication by endocrinologist is reported.
  Age for each patient was calculated by subtracting the year of birth from the year of registration (i.e. Year of registration - Year of birth). Year of registration was defined as the year the patients where initiated on T2D medication.
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: Patients of the prescribed patient set (PPS) who were initiated on type 2 diabetes (T2D) medication by endocrinologist. PPS included all patients fulfilling inclusion and exclusion criteria who have received a first prescription of a respective T2D medication and whose documentation was electronically signed by the physician.
Measure: Mean (Standard Deviation); unit: Years
Groups:
- Patients Initiated on Empagliflozin by Endocrinologist: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on empagliflozin between September 2018 and December 2018 (study index date 1) by endocrinologist.
- Patients Initiated on DPP4i by Endocrinologist: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on dipeptidyl peptidase 4 inhibitor (DPP4i) between September 2018 and December 2018 (study index date 1) by endocrinologist.
- Patients Initiated on GLP-1 RA by Endocrinologist: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on glucagon-like peptide-1 receptor agonist (GLP-1 RA) between September 2018 and December 2018 (study index date 1) by endocrinologist.
- Patients Initiated on Other SGLT2i by Endocrinologist: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on other sodium dependent glucose transporter inhibitor (SGLT2i) between September 2018 and December 2018 (study index date 1) by endocrinologist.
Arm/Group | Patients Initiated on Empagliflozin by Endocrinologist | Patients Initiated on DPP4i by Endocrinologist | Patients Initiated on GLP-1 RA by Endocrinologist | Patients Initiated on Other SGLT2i by Endocrinologist
Number analyzed (Participants) | 815 | 504 | 89 | 244
Years | 61.5 (9.7) | 65.3 (10.4) | 55.8 (10.5) | 62.0 (9.2)
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Endocrinologist vs Patients Initiated on DPP4i by Endocrinologist vs Patients Initiated on GLP-1 RA by Endocrinologist vs Patients Initiated on Other SGLT2i by Endocrinologist; Test type: Other; p < .0001, Kruskal-Wallis

5. Primary Outcome: Baseline Characteristic: Number of Patients in Each Category of Gender According to Type 2 Diabetes (T2D) Medication for the Patients Who Were Initiated on T2D Medication by Endocrinologist
Description: Baseline characteristic: Number of patients in each category of gender according to type 2 diabetes (T2D) medication for the patients who were initiated on T2D medication by endocrinologist is reported.
  The reported categories of gender are:
  * Female
  * Male
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on Empagliflozin by Endocrinologist | Patients Initiated on DPP4i by Endocrinologist | Patients Initiated on GLP-1 RA by Endocrinologist | Patients Initiated on Other SGLT2i by Endocrinologist
Number analyzed (Participants) | 815 | 504 | 89 | 244
Participants
  Female | 432 | 334 | 37 | 140
  Male | 383 | 170 | 52 | 104
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Endocrinologist vs Patients Initiated on DPP4i by Endocrinologist vs Patients Initiated on GLP-1 RA by Endocrinologist vs Patients Initiated on Other SGLT2i by Endocrinologist; Test type: Other; p < .0001, Chi-squared

6. Primary Outcome: Baseline Characteristic: Body Mass Index (BMI) According to Type 2 Diabetes (T2D) Medication for the Patients Who Were Initiated on T2D Medication by Endocrinologist
Description: Baseline characteristic: Body mass index (BMI) according to type 2 diabetes (T2D) medication for the patients who were initiated on T2D medication by endocrinologist is reported.
  Body mass index (BMI) is weight in kilograms divided by height in meters squared (kilogram/meter^2 (kg/m^2)).
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: kilogram/meter^2 (kg/m^2)
Arm/Group | Patients Initiated on Empagliflozin by Endocrinologist | Patients Initiated on DPP4i by Endocrinologist | Patients Initiated on GLP-1 RA by Endocrinologist | Patients Initiated on Other SGLT2i by Endocrinologist
Number analyzed (Participants) | 815 | 504 | 89 | 244
kilogram/meter^2 (kg/m^2) | 33.3 (5.4) | 31.3 (5.2) | 36.7 (5.9) | 34.3 (5.8)
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Endocrinologist vs Patients Initiated on DPP4i by Endocrinologist vs Patients Initiated on GLP-1 RA by Endocrinologist vs Patients Initiated on Other SGLT2i by Endocrinologist; Test type: Other; p < .0001, Kruskal-Wallis

7. Primary Outcome: Baseline Characteristic: Number of Patients in Each Category of Race According to Type 2 Diabetes (T2D) Medication for the Patients Who Were Initiated on T2D Medication by Endocrinologist
Description: Baseline characteristic: Number of patients in each category of race according to type 2 diabetes (T2D) medication for the patients who were initiated on T2D medication by endocrinologist is reported.
  The reported categories of race are:
  * Black
  * Non-black
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on Empagliflozin by Endocrinologist | Patients Initiated on DPP4i by Endocrinologist | Patients Initiated on GLP-1 RA by Endocrinologist | Patients Initiated on Other SGLT2i by Endocrinologist
Number analyzed (Participants) | 815 | 504 | 89 | 244
Participants
  Black | 10 | 7 | 1 | 5
  Non-black | 805 | 497 | 88 | 239
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Endocrinologist vs Patients Initiated on DPP4i by Endocrinologist vs Patients Initiated on GLP-1 RA by Endocrinologist vs Patients Initiated on Other SGLT2i by Endocrinologist; Test type: Other; p = 0.8071, Chi-squared
Statistical Analysis 2: Comparison: Patients Initiated on Empagliflozin by Endocrinologist vs Patients Initiated on DPP4i by Endocrinologist vs Patients Initiated on GLP-1 RA by Endocrinologist vs Patients Initiated on Other SGLT2i by Endocrinologist; Test type: Other; p = 0.7640, Fisher Exact

8. Primary Outcome: Baseline Characteristic: Age According to Type 2 Diabetes (T2D) Medication for the Patients Who Were Initiated on T2D Medication by Diabetologist
Description: Baseline characteristic: Age according to type 2 diabetes (T2D) medication for the patients who were initiated on T2D medication by diabetologist is reported.
  Age for each patient was calculated by subtracting the year of birth from the year of registration (i.e. Year of registration - Year of birth). Year of registration was defined as the year the patients where initiated on T2D medication.
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: Patients of the prescribed patient set (PPS) who were initiated on type 2 diabetes (T2D) medication by diabetologist. PPS included all patients fulfilling inclusion and exclusion criteria who have received a first prescription of a respective T2D medication and whose documentation was electronically signed by the physician.
Measure: Mean (Standard Deviation); unit: Years
Groups:
- Patients Initiated on Empagliflozin by Diabetologist: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on empagliflozin between September 2018 and December 2018 (study index date 1) by diabetologist.
- Patients Initiated on DPP4i by Diabetologist: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on dipeptidyl peptidase 4 inhibitor (DPP4i) between September 2018 and December 2018 (study index date 1) by diabetologist.
- Patients Initiated on GLP-1 RA by Diabetologist: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on glucagon-like peptide-1 receptor agonist (GLP-1 RA) between September 2018 and December 2018 (study index date 1)by diabetologist.
- Patients Initiated on Other SGLT2i by Diabetologist: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on other sodium dependent glucose transporter inhibitor (SGLT2i) between September 2018 and December 2018 (study index date 1) by diabetologist.
Arm/Group | Patients Initiated on Empagliflozin by Diabetologist | Patients Initiated on DPP4i by Diabetologist | Patients Initiated on GLP-1 RA by Diabetologist | Patients Initiated on Other SGLT2i by Diabetologist
Number analyzed (Participants) | 1073 | 624 | 271 | 333
Years | 63.0 (9.4) | 67.2 (11.0) | 59.2 (10.8) | 62.3 (9.2)
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Diabetologist vs Patients Initiated on DPP4i by Diabetologist vs Patients Initiated on GLP-1 RA by Diabetologist vs Patients Initiated on Other SGLT2i by Diabetologist; Test type: Other; p < .0001, Kruskal-Wallis

9. Primary Outcome: Baseline Characteristic: Number of Patients in Each Category of Gender According to Type 2 Diabetes (T2D) Medication for the Patients Who Were Initiated on T2D Medication by Diabetologist
Description: Baseline characteristic: Number of patients in each category of gender according to type 2 diabetes (T2D) medication for the patients who were initiated on T2D medication by diabetologist is reported.
  The reported categories of gender are:
  * Female
  * Male
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Groups:
- Patients Initiated on GLP-1 RA by Diabetologist: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on glucagon-like peptide-1 receptor agonist (GLP-1 RA) between September 2018 and December 2018 (study index date 1) by diabetologist.
Arm/Group | Patients Initiated on Empagliflozin by Diabetologist | Patients Initiated on DPP4i by Diabetologist | Patients Initiated on GLP-1 RA by Diabetologist | Patients Initiated on Other SGLT2i by Diabetologist
Number analyzed (Participants) | 1073 | 624 | 271 | 333
Participants
  Female | 433 | 297 | 135 | 140
  Male | 640 | 327 | 136 | 193
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Diabetologist vs Patients Initiated on DPP4i by Diabetologist vs Patients Initiated on GLP-1 RA by Diabetologist vs Patients Initiated on Other SGLT2i by Diabetologist; Test type: Other; p = 0.0042, Chi-squared

10. Primary Outcome: Body Mass Index (BMI) According to Type 2 Diabetes (T2D) Medication for the Patients Who Were Initiated on T2D Medication by Diabetologist
Description: Baseline characteristic: Body mass index (BMI) according to type 2 diabetes (T2D) medication for the patients who were initiated on T2D medication by diabetologist is reported.
  Body mass index (BMI) is weight in kilograms divided by height in meters squared (kilogram/meter^2 (kg/m^2)).
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: kilogram/meter^2 (kg/m^2)
Arm/Group | Patients Initiated on Empagliflozin by Diabetologist | Patients Initiated on DPP4i by Diabetologist | Patients Initiated on GLP-1 RA by Diabetologist | Patients Initiated on Other SGLT2i by Diabetologist
Number analyzed (Participants) | 1073 | 624 | 271 | 333
kilogram/meter^2 (kg/m^2) | 33.3 (5.9) | 31.0 (5.4) | 36.2 (6.7) | 32.8 (5.3)
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Diabetologist vs Patients Initiated on DPP4i by Diabetologist vs Patients Initiated on GLP-1 RA by Diabetologist vs Patients Initiated on Other SGLT2i by Diabetologist; Test type: Other; p < .0001, Kruskal-Wallis

11. Primary Outcome: Baseline Characteristic: Number of Patients in Each Category of Race According to Type 2 Diabetes (T2D) Medication for the Patients Who Were Initiated on T2D Medication by Diabetologist
Description: Baseline characteristic: Number of patients in each category of race according to type 2 diabetes (T2D) medication for the patients who were initiated on T2D medication by diabetologist is reported.
  The reported categories of race are:
  * Black
  * Non-black
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on Empagliflozin by Diabetologist | Patients Initiated on DPP4i by Diabetologist | Patients Initiated on GLP-1 RA by Diabetologist | Patients Initiated on Other SGLT2i by Diabetologist
Number analyzed (Participants) | 1073 | 624 | 271 | 333
Participants
  Black | 3 | 0 | 1 | 0
  Non-black | 1070 | 624 | 270 | 333
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Diabetologist vs Patients Initiated on DPP4i by Diabetologist vs Patients Initiated on GLP-1 RA by Diabetologist vs Patients Initiated on Other SGLT2i by Diabetologist; Test type: Other; p = 0.3990, Chi-squared
Statistical Analysis 2: Comparison: Patients Initiated on Empagliflozin by Diabetologist vs Patients Initiated on DPP4i by Diabetologist vs Patients Initiated on GLP-1 RA by Diabetologist vs Patients Initiated on Other SGLT2i by Diabetologist; Test type: Other; p = 0.3842, Fisher Exact

12. Primary Outcome: Baseline Characteristic: Age According to Type 2 Diabetes (T2D) Medication for the Patients Who Were Initiated on T2D Medication by Cardiologist
Description: Baseline characteristic: Age according to type 2 diabetes (T2D) medication for the patients who were initiated on T2D medication by cardiologist is reported.
  Age for each patient was calculated by subtracting the year of birth from the year of registration (i.e. Year of registration - Year of birth). Year of registration was defined as the year the patients where initiated on T2D medication.
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: Patients of the prescribed patient set (PPS) who were initiated on type 2 diabetes (T2D) medication by cardiologist. PPS included all patients fulfilling inclusion and exclusion criteria who have received a first prescription of a respective T2D medication and whose documentation was electronically signed by the physician.
Measure: Mean (Standard Deviation); unit: Years
Groups:
- Patients Initiated on Empagliflozin by Cardiologist: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on empagliflozin between September 2018 and December 2018 (study index date 1) by cardiologist.
- Patients Initiated on DPP4i by Cardiologist: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on dipeptidyl peptidase 4 inhibitor (DPP4i) between September 2018 and December 2018 (study index date 1) by cardiologist.
- Patients Initiated on GLP-1 RA by Cardiologist: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on glucagon-like peptide-1 receptor agonist (GLP-1 RA) between September 2018 and December 2018 (study index date 1) by cardiologist.
- Patients Initiated on Other SGLT2i by Cardiologist: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on other sodium dependent glucose transporter inhibitor (SGLT2i) between September 2018 and December 2018 (study index date 1) by cardiologist.
Arm/Group | Patients Initiated on Empagliflozin by Cardiologist | Patients Initiated on DPP4i by Cardiologist | Patients Initiated on GLP-1 RA by Cardiologist | Patients Initiated on Other SGLT2i by Cardiologist
Number analyzed (Participants) | 78 | 16 | 1 | 7
Years | 64.4 (8.4) | 70.9 (9.5) | 54.0 | 65.0 (9.4)
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Cardiologist vs Patients Initiated on DPP4i by Cardiologist vs Patients Initiated on GLP-1 RA by Cardiologist vs Patients Initiated on Other SGLT2i by Cardiologist; Test type: Other; p = 0.0605, Kruskal-Wallis

13. Primary Outcome: Baseline Characteristic: Number of Patients in Each Category of Gender According to Type 2 Diabetes (T2D) Medication for the Patients Who Were Initiated on T2D Medication by Cardiologist
Description: Baseline characteristic: Number of patients in each category of gender according to type 2 diabetes (T2D) medication for the patients who were initiated on T2D medication by cardiologist is reported.
  The reported categories of gender are:
  * Female
  * Male
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on Empagliflozin by Cardiologist | Patients Initiated on DPP4i by Cardiologist | Patients Initiated on GLP-1 RA by Cardiologist | Patients Initiated on Other SGLT2i by Cardiologist
Number analyzed (Participants) | 78 | 16 | 1 | 7
Participants
  Female | 35 | 8 | 0 | 2
  Male | 43 | 8 | 1 | 5
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Cardiologist vs Patients Initiated on DPP4i by Cardiologist vs Patients Initiated on GLP-1 RA by Cardiologist vs Patients Initiated on Other SGLT2i by Cardiologist; Test type: Other; p = 0.6329, Chi-squared
Statistical Analysis 2: Comparison: Patients Initiated on Empagliflozin by Cardiologist vs Patients Initiated on DPP4i by Cardiologist vs Patients Initiated on GLP-1 RA by Cardiologist vs Patients Initiated on Other SGLT2i by Cardiologist; Test type: Other; p = 0.7181, Fisher Exact

14. Primary Outcome: Body Mass Index (BMI) According to Type 2 Diabetes (T2D) Medication for the Patients Who Were Initiated on T2D Medication by Cardiologist
Description: Baseline characteristic: Body mass index (BMI) according to type 2 diabetes (T2D) medication for the patients who were initiated on T2D medication by cardiologist is reported.
  Body mass index (BMI) is weight in kilograms divided by height in meters squared (kilogram/meter^2 (kg/m^2)).
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: kilogram/meter^2 (kg/m^2)
Groups:
- Patients Initiated on DPP4i by Cardiologist: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) with dipeptidyl peptidase 4 inhibitor (DPP4i) between September 2018 and December 2018 (study index date 1) by cardiologist.
Arm/Group | Patients Initiated on Empagliflozin by Cardiologist | Patients Initiated on DPP4i by Cardiologist | Patients Initiated on GLP-1 RA by Cardiologist | Patients Initiated on Other SGLT2i by Cardiologist
Number analyzed (Participants) | 78 | 16 | 1 | 7
kilogram/meter^2 (kg/m^2) | 30.8 (4.6) | 29.9 (4.2) | 25.8 | 30.7 (2.3)
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Cardiologist vs Patients Initiated on DPP4i by Cardiologist vs Patients Initiated on GLP-1 RA by Cardiologist vs Patients Initiated on Other SGLT2i by Cardiologist; Test type: Other; p = 0.5233, Kruskal-Wallis

15. Primary Outcome: Baseline Characteristic: Number of Patients in Each Category of Race According to Type 2 Diabetes (T2D) Medication for the Patients Who Were Initiated on T2D Medication by Cardiologist
Description: Baseline characteristic: Number of patients in each category of race according to type 2 diabetes (T2D) medication for the patients who were initiated on T2D medication by cardiologist is reported.
  The reported categories of race are:
  * Black
  * Non-black
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on Empagliflozin by Cardiologist | Patients Initiated on DPP4i by Cardiologist | Patients Initiated on GLP-1 RA by Cardiologist | Patients Initiated on Other SGLT2i by Cardiologist
Number analyzed (Participants) | 78 | 16 | 1 | 7
Participants
  Black | 0 | 0 | 0 | 0
  Non-black | 78 | 16 | 1 | 7

16. Primary Outcome: Time Since Diagnosis of Type 2 Diabetes (T2D) According to T2D Medication for the Patients Who Were Initiated on T2D Medication by Endocrinologist
Description: Time since diagnosis of type 2 diabetes (T2D) according to T2D medication for the patients who were initiated on T2D medication by endocrinologist is reported.
  Time since diagnosis of T2D (years) was calculated by subtracting the year of T2D diagnosis from the year of registration. Year of registration was defined as the year patients where initiated on T2D medication.
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Patients Initiated on Empagliflozin by Endocrinologist | Patients Initiated on DPP4i by Endocrinologist | Patients Initiated on GLP-1 RA by Endocrinologist | Patients Initiated on Other SGLT2i by Endocrinologist
Number analyzed (Participants) | 815 | 504 | 89 | 244
Years | 9.1 (6.6) | 9.1 (6.6) | 9.2 (6.9) | 9.8 (6.7)
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Endocrinologist vs Patients Initiated on DPP4i by Endocrinologist vs Patients Initiated on GLP-1 RA by Endocrinologist vs Patients Initiated on Other SGLT2i by Endocrinologist; Test type: Other; p = 0.3662, Kruskal-Wallis

17. Primary Outcome: Time Since Diagnosis of Type 2 Diabetes (T2D) According to T2D Medication for the Patients Who Were Initiated on T2D Medication by Diabetologist
Description: Time since diagnosis of type 2 diabetes (T2D) according to T2D medication for the patients who were initiated on T2D medication by diabetologist is reported.
  Time since diagnosis of T2D (years) was calculated by subtracting the year of T2D diagnosis from the year of registration. Year of registration was defined as the year patients where initiated on T2D medication.
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Years
Groups:
- Patients Initiated on Other SGLT2i by Diabetologist: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who on other sodium dependent glucose transporter inhibitor (SGLT2i) between September 2018 and December 2018 (study index date 1) by diabetologist.
Arm/Group | Patients Initiated on Empagliflozin by Diabetologist | Patients Initiated on DPP4i by Diabetologist | Patients Initiated on GLP-1 RA by Diabetologist | Patients Initiated on Other SGLT2i by Diabetologist
Number analyzed (Participants) | 1073 | 624 | 271 | 333
Years | 10.7 (7.3) | 10.4 (7.3) | 10.1 (6.6) | 10.1 (6.8)
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Diabetologist vs Patients Initiated on DPP4i by Diabetologist vs Patients Initiated on GLP-1 RA by Diabetologist vs Patients Initiated on Other SGLT2i by Diabetologist; Test type: Other; p = 0.5110, Kruskal-Wallis

18. Primary Outcome: Time Since Diagnosis of Type 2 Diabetes (T2D) According to T2D Medication for the Patients Who Were Initiated on T2D Medication by Cardiologist
Description: Time since diagnosis of type 2 diabetes (T2D) according to T2D medication for the patients who were initiated on T2D medication by cardiologist is reported.
  Time since diagnosis of T2D (years) was calculated by subtracting the year of T2D diagnosis from the year of registration. Year of registration was defined as the year patients where initiated on T2D medication.
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Patients Initiated on Empagliflozin by Cardiologist | Patients Initiated on DPP4i by Cardiologist | Patients Initiated on GLP-1 RA by Cardiologist | Patients Initiated on Other SGLT2i by Cardiologist
Number analyzed (Participants) | 78 | 16 | 1 | 7
Years | 6.7 (4.0) | 9.7 (5.7) | 6.0 | 10.9 (6.5)
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Cardiologist vs Patients Initiated on DPP4i by Cardiologist vs Patients Initiated on GLP-1 RA by Cardiologist vs Patients Initiated on Other SGLT2i by Cardiologist; Test type: Other; p = 0.0921, Kruskal-Wallis

19. Primary Outcome: Clinical Parameter Relevant for Type 2 Diabetes (T2D): Percentage of Glycosylated Hemoglobin (HbA1c [%]) According to T2D Medication for the Patients Who Were Initiated on T2D Medication by Endocrinologist
Description: Clinical parameter relevant for Type 2 Diabetes (T2D): Percentage of glycosylated hemoglobin (HbA1c [%]) according to T2D medication for the patients who were initiated on T2D medication by endocrinologist is reported.
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: Patients of the prescribed patient set (PPS) who were initiated on type 2 diabetes (T2D) medication by endocrinologist. PPS included all patients fulfilling inclusion and exclusion criteria who have received a first prescription of a respective T2D medication and whose documentation was electronically signed by the physician. Only participants with non-missing results are reported.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Patients Initiated on Empagliflozin by Endocrinologist | Patients Initiated on DPP4i by Endocrinologist | Patients Initiated on GLP-1 RA by Endocrinologist | Patients Initiated on Other SGLT2i by Endocrinologist
Number analyzed (Participants) | 802 | 477 | 85 | 235
percentage of glycosylated hemoglobin | 8.5 (1.4) | 8.1 (1.2) | 8.2 (1.1) | 8.5 (1.3)
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Endocrinologist vs Patients Initiated on DPP4i by Endocrinologist vs Patients Initiated on GLP-1 RA by Endocrinologist vs Patients Initiated on Other SGLT2i by Endocrinologist; Test type: Other; p < .0001, Kruskal-Wallis

20. Primary Outcome: Clinical Parameter Relevant for T2D: Number of Patients in Each Category of Percentage of Glycosylated Hemoglobin (HbA1c) According to T2D Medication for the Patients Who Were Initiated on T2D Medication by Endocrinologist
Description: Clinical parameter relevant for Type 2 Diabetes (T2D): Number of patients in each category of percentage of glycosylated hemoglobin (HbA1c) according to T2D medication for the patients who were initiated on T2D medication by endocrinologist is reported.
  The reported categories of percentage (%) of glycosylated hemoglobin are:
  * <8.5%
  * ≥8.5%
  * Missing
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on Empagliflozin by Endocrinologist | Patients Initiated on DPP4i by Endocrinologist | Patients Initiated on GLP-1 RA by Endocrinologist | Patients Initiated on Other SGLT2i by Endocrinologist
Number analyzed (Participants) | 815 | 504 | 89 | 244
Participants
  <8.5% | 453 | 339 | 56 | 138
  ≥8.5% | 349 | 138 | 29 | 97
  Missing | 13 | 27 | 4 | 9
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Endocrinologist vs Patients Initiated on DPP4i by Endocrinologist vs Patients Initiated on GLP-1 RA by Endocrinologist vs Patients Initiated on Other SGLT2i by Endocrinologist; Test type: Other; p < .0001, Chi-squared

21. Primary Outcome: Clinical Parameter Relevant for Type 2 Diabetes (T2D): Percentage of Glycosylated Hemoglobin (HbA1c [%]) According to T2D Medication for the Patients Who Were Initiated on T2D Medication by Diabetologist
Description: Clinical parameter relevant for type 2 diabetes (T2D): Percentage of glycosylated hemoglobin (HbA1c [%]) according to T2D medication for the patients who were initiated on T2D medication by diabetologist is reported.
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: Patients of the prescribed patient set (PPS) who were initiated on type by diabetologist. PPS included all patients fulfilling inclusion and exclusion criteria who have received a first prescription of a respective T2D medication and whose documentation was electronically signed by the physician. Only participants with non-missing results are reported.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Patients Initiated on Empagliflozin by Diabetologist | Patients Initiated on DPP4i by Diabetologist | Patients Initiated on GLP-1 RA by Diabetologist | Patients Initiated on Other SGLT2i by Diabetologist
Number analyzed (Participants) | 920 | 576 | 257 | 297
percentage of glycosylated hemoglobin | 8.2 (1.3) | 7.9 (1.4) | 8.4 (1.2) | 8.6 (1.6)
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Diabetologist vs Patients Initiated on DPP4i by Diabetologist vs Patients Initiated on GLP-1 RA by Diabetologist vs Patients Initiated on Other SGLT2i by Diabetologist; Test type: Other; p < .0001, Kruskal-Wallis

22. Primary Outcome: Clinical Parameter Relevant for Type 2 Diabetes (T2D): Number of Patients in Each Category of Percentage of Glycosylated Hemoglobin (HbA1c) According to T2D Medication for the Patients Who Were Initiated on T2D Medication by Diabetologist
Description: Clinical parameter relevant for type 2 diabetes (T2D): Number of patients in each category of percentage of glycosylated hemoglobin (HbA1c) according to T2D medication for the patients who were initiated on T2D medication by diabetologist is reported.
  The reported categories of percentage of glycosylated hemoglobin are:
  * <8.5%
  * ≥8.5%
  * Missing
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on Empagliflozin by Diabetologist | Patients Initiated on DPP4i by Diabetologist | Patients Initiated on GLP-1 RA by Diabetologist | Patients Initiated on Other SGLT2i by Diabetologist
Number analyzed (Participants) | 1073 | 624 | 271 | 333
Participants
  <8.5% | 642 | 453 | 162 | 183
  ≥8.5% | 278 | 123 | 95 | 114
  Missing | 153 | 48 | 14 | 36
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Diabetologist vs Patients Initiated on DPP4i by Diabetologist vs Patients Initiated on GLP-1 RA by Diabetologist vs Patients Initiated on Other SGLT2i by Diabetologist; Test type: Other; p < .0001, Chi-squared

23. Primary Outcome: Clinical Parameter Relevant for Type 2 Diabetes (T2D): Percentage of Glycosylated Hemoglobin (HbA1c [%]) According to T2D Medication for the Patients Who Were Initiated on T2D Medication by Cardiologist
Description: Clinical parameter relevant for type 2 diabetes (T2D): Percentage of glycosylated hemoglobin (HbA1c [%]) according to T2D medication for the patients who were initiated on T2D medication by cardiologist is reported.
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: Patients of the prescribed patient set (PPS) who were initiated on type 2 diabetes (T2D) medication by cardiologist. PPS included all patients fulfilling inclusion and exclusion criteria who have received a first prescription of a respective T2D medication and whose documentation was electronically signed by the physician. Only patients with non-missing values are reported.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Groups:
- Patients Initiated on DPP4i by Cardiologist: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on dipeptidyl peptidase 4 inhibitor (DPP4i) between September 2018 and by cardiologist.
Arm/Group | Patients Initiated on Empagliflozin by Cardiologist | Patients Initiated on DPP4i by Cardiologist | Patients Initiated on GLP-1 RA by Cardiologist | Patients Initiated on Other SGLT2i by Cardiologist
Number analyzed (Participants) | 50 | 15 | 1 | 5
percentage of glycosylated hemoglobin | 7.9 (1.1) | 8.1 (1.1) | 7.4 | 8.5 (0.7)
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Cardiologist vs Patients Initiated on DPP4i by Cardiologist vs Patients Initiated on GLP-1 RA by Cardiologist vs Patients Initiated on Other SGLT2i by Cardiologist; Test type: Other; p = 0.3201, Kruskal-Wallis

24. Primary Outcome: Clinical Parameter Relevant for Type 2 Diabetes (T2D): Number of Patients in Each Category of Percentage of Glycosylated Hemoglobin (HbA1c) According to T2D Medication for the Patients Who Were Initiated on T2D Medication by Cardiologist
Description: Clinical parameter relevant for type 2 diabetes (T2D): Number of patients in each category of percentage of glycosylated hemoglobin (HbA1c) according to T2D medication for the patients who were initiated on T2D medication by cardiologist is reported.
  The reported categories of percentage of glycosylated hemoglobin are:
  * <8.5%
  * ≥8.5%
  * Missing
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on Empagliflozin by Cardiologist | Patients Initiated on DPP4i by Cardiologist | Patients Initiated on GLP-1 RA by Cardiologist | Patients Initiated on Other SGLT2i by Cardiologist
Number analyzed (Participants) | 78 | 16 | 1 | 7
Participants
  <8.5% | 36 | 11 | 1 | 3
  ≥8.5% | 14 | 4 | 0 | 2
  Missing | 28 | 1 | 0 | 2
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Cardiologist vs Patients Initiated on DPP4i by Cardiologist vs Patients Initiated on GLP-1 RA by Cardiologist vs Patients Initiated on Other SGLT2i by Cardiologist; Test type: Other; p = 0.3288, Chi-squared
Statistical Analysis 2: Comparison: Patients Initiated on Empagliflozin by Cardiologist vs Patients Initiated on DPP4i by Cardiologist vs Patients Initiated on GLP-1 RA by Cardiologist vs Patients Initiated on Other SGLT2i by Cardiologist; Test type: Other; p = 0.1710, Fisher Exact

25. Primary Outcome: 10-year Risk for Fatal Cardiovascular Disease (CVD) According to Type 2 Diabetes (T2D) Medication for the Patients Who Were Initiated on T2D Medication by Endocrinologist
Description: 10-year risk for fatal cardiovascular disease (CVD) according to type 2 diabetes (T2D) medication for the patients who were initiated on T2D medication by endocrinologist is reported.
  10-year risk for fatal CVD was calculated according to the applying Systematic COronary Risk Evaluation (SCORE) Risk Chart (European Society of Cardiology) which takes into account patient´s age, gender, systolic blood pressure, smoking status, and total cholesterol value at index date 1. SCORE Risk Chart takes values from from 0% to 100%. SCORE Risk Chart values from 5% and upwards indicate a high 10-year risk for a fatal cardiovascular event.
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: Patients of the prescribed patient set (PPS) who were initiated on type 2 diabetes (T2D) medication by endocrinologist. PPS included all patients fulfilling inclusion and exclusion criteria who have received a first prescription of a respective T2D medication and whose documentation was electronically signed by the physician. Only patients with non-missing results are reported.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Patients Initiated on Empagliflozin by Endocrinologist | Patients Initiated on DPP4i by Endocrinologist | Patients Initiated on GLP-1 RA by Endocrinologist | Patients Initiated on Other SGLT2i by Endocrinologist
Number analyzed (Participants) | 615 | 403 | 62 | 179
Score on a scale | 6.4 (5.7) | 5.6 (4.7) | 4.3 (3.7) | 6.0 (5.7)
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Endocrinologist vs Patients Initiated on DPP4i by Endocrinologist vs Patients Initiated on GLP-1 RA by Endocrinologist vs Patients Initiated on Other SGLT2i by Endocrinologist; Test type: Other; p = 0.0130, Kruskal-Wallis

26. Primary Outcome: 10-year Risk for Fatal Cardiovascular Disease (CVD) According to Type 2 Diabetes (T2D) Medication for the Patients Who Were Initiated on T2D Medication by Diabetologist
Description: 10-year risk for fatal cardiovascular disease (CVD) according to type 2 diabetes (T2D) medication for the patients who were initiated on T2D medication by diabetologist is reported.
  10-year risk for fatal CVD was calculated according to the applying Systematic COronary Risk Evaluation (SCORE) Risk Chart (European Society of Cardiology) which takes into account patient´s age, gender, systolic blood pressure, smoking status, and total cholesterol value at index date 1. SCORE Risk Chart takes values from from 0% to 100%. SCORE Risk Chart values from 5% and upwards indicate a high 10-year risk for a fatal cardiovascular event.
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: Patients of the prescribed patient set (PPS) who were initiated on type 2 diabetes (T2D) medication by diabetologist. PPS included all patients fulfilling inclusion and exclusion criteria who have received a first prescription of a respective T2D medication and whose documentation was electronically signed by the physician. Only patients with non-missing results are reported.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Patients Initiated on Empagliflozin by Diabetologist | Patients Initiated on DPP4i by Diabetologist | Patients Initiated on GLP-1 RA by Diabetologist | Patients Initiated on Other SGLT2i by Diabetologist
Number analyzed (Participants) | 609 | 355 | 155 | 164
Score on a scale | 7.0 (5.5) | 7.0 (5.9) | 5.4 (4.7) | 6.5 (5.1)
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Diabetologist vs Patients Initiated on DPP4i by Diabetologist vs Patients Initiated on GLP-1 RA by Diabetologist vs Patients Initiated on Other SGLT2i by Diabetologist; Test type: Other; p = 0.0026, Kruskal-Wallis

27. Primary Outcome: 10-year Risk for Fatal Cardiovascular Disease (CVD) According to Type 2 Diabetes (T2D) Medication for the Patients Who Were Initiated on T2D Medication by Cardiologist
Description: 10-year risk for fatal cardiovascular disease (CVD) according to type 2 diabetes (T2D) medication for the patients who were initiated on T2D medication by cardiologist is reported.
  10-year risk for fatal CVD was calculated according to the applying Systematic COronary Risk Evaluation (SCORE) Risk Chart (European Society of Cardiology) which takes into account patient´s age, gender, systolic blood pressure, smoking status, and total cholesterol value at index date 1. SCORE Risk Chart takes values from from 0% to 100%. SCORE Risk Chart values from 5% and upwards indicate a high 10-year risk for a fatal cardiovascular event.
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: Patients of the prescribed patient set (PPS) who were initiated on type 2 diabetes (T2D) medication by cardiologist. PPS included all patients fulfilling inclusion and exclusion criteria who have received a first prescription of a respective T2D medication and whose documentation was electronically signed by the physician. Only patients with non-missing results are reported.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Patients Initiated on DPP4i by Cardiologist: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who on dipeptidyl peptidase 4 inhibitor (DPP4i) between September 2018 and December 2018 (study index date 1) by cardiologist.
Arm/Group | Patients Initiated on Empagliflozin by Cardiologist | Patients Initiated on DPP4i by Cardiologist | Patients Initiated on GLP-1 RA by Cardiologist | Patients Initiated on Other SGLT2i by Cardiologist
Number analyzed (Participants) | 54 | 11 | 1 | 5
Score on a scale | 8.9 (7.7) | 9.4 (7.8) | 5.0 | 3.8 (2.3)
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Cardiologist vs Patients Initiated on DPP4i by Cardiologist vs Patients Initiated on GLP-1 RA by Cardiologist vs Patients Initiated on Other SGLT2i by Cardiologist; Test type: Other; p = 0.3978, Kruskal-Wallis

28. Primary Outcome: Number of Patients Per Type of Medical Specialty of Other Physicians Involved in Treatment Decision According to Type 2 Diabetes (T2D) Medication for the Patients Who Were Initiated on T2D Medication by Endocrinologist
Description: Number of patients per type of medical specialty of other physicians involved in treatment decision according to type 2 diabetes (T2D) medication for the patients who were initiated on T2D medication by endocrinologist is reported.
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on Empagliflozin by Endocrinologist | Patients Initiated on DPP4i by Endocrinologist | Patients Initiated on GLP-1 RA by Endocrinologist | Patients Initiated on Other SGLT2i by Endocrinologist
Number analyzed (Participants) | 815 | 504 | 89 | 244
Participants
  Other endocrinologist | 56 | 36 | 1 | 11
  Diabetologist | 0 | 0 | 0 | 0
  Cardiologist | 81 | 25 | 7 | 19
  Nephrologist | 8 | 8 | 2 | 0
  General practitioner | 46 | 33 | 7 | 12
  Others | 3 | 5 | 3 | 1
  None | 697 | 439 | 76 | 209
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Endocrinologist vs Patients Initiated on DPP4i by Endocrinologist vs Patients Initiated on GLP-1 RA by Endocrinologist vs Patients Initiated on Other SGLT2i by Endocrinologist; Test type: Other; p = 0.0055, Chi-squared
Statistical Analysis 2: Comparison: Patients Initiated on Empagliflozin by Endocrinologist vs Patients Initiated on DPP4i by Endocrinologist vs Patients Initiated on GLP-1 RA by Endocrinologist vs Patients Initiated on Other SGLT2i by Endocrinologist; Test type: Other; p = 0.0041, Fisher Exact

29. Primary Outcome: Number of Patients Per Type of Medical Specialty of Other Physicians Involved in Treatment Decision According to Type 2 Diabetes (T2D) Medication for the Patients Who Were Initiated on T2D Medication by Diabetologist
Description: Number of patients per type of medical specialty of other physicians involved in treatment decision according to type 2 diabetes (T2D) medication for the patients who were initiated on T2D medication by diabetologist is reported.
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on Empagliflozin by Diabetologist | Patients Initiated on DPP4i by Diabetologist | Patients Initiated on GLP-1 RA by Diabetologist | Patients Initiated on Other SGLT2i by Diabetologist
Number analyzed (Participants) | 1073 | 624 | 271 | 333
Participants
  Endocrinologist | 3 | 0 | 0 | 0
  Other diabetologist | 74 | 35 | 11 | 24
  Cardiologist | 35 | 2 | 2 | 3
  Nephrologist | 1 | 5 | 0 | 0
  General practitioner | 25 | 6 | 1 | 7
  Others | 0 | 1 | 0 | 1
  None | 953 | 577 | 257 | 300
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Diabetologist vs Patients Initiated on DPP4i by Diabetologist vs Patients Initiated on GLP-1 RA by Diabetologist vs Patients Initiated on Other SGLT2i by Diabetologist; Test type: Other; p < .0001, Chi-squared

30. Primary Outcome: Number of Patients Per Type of Medical Specialty of Other Physicians Involved in Treatment Decision According to Type 2 Diabetes (T2D) Medication for the Patients Who Were Initiated on T2D Medication by Cardiologist
Description: Number of patients per type of medical specialty of other physicians involved in treatment decision according to type 2 diabetes (T2D) medication for the patients who were initiated on T2D medication by cardiologist is reported.
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on Empagliflozin by Cardiologist | Patients Initiated on DPP4i by Cardiologist | Patients Initiated on GLP-1 RA by Cardiologist | Patients Initiated on Other SGLT2i by Cardiologist
Number analyzed (Participants) | 78 | 16 | 1 | 7
Participants
  Endocrinologist | 19 | 0 | 0 | 0
  Diabetologist | 10 | 1 | 0 | 0
  Other cardiologist | 4 | 0 | 0 | 0
  Nephrologist | 1 | 3 | 0 | 0
  General practitioner | 0 | 0 | 0 | 0
  Others | 0 | 0 | 0 | 0
  None | 45 | 12 | 1 | 7
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Cardiologist vs Patients Initiated on DPP4i by Cardiologist vs Patients Initiated on GLP-1 RA by Cardiologist vs Patients Initiated on Other SGLT2i by Cardiologist; Test type: Other; p = 0.0399, Chi-squared
Statistical Analysis 2: Comparison: Patients Initiated on Empagliflozin by Cardiologist vs Patients Initiated on DPP4i by Cardiologist vs Patients Initiated on GLP-1 RA by Cardiologist vs Patients Initiated on Other SGLT2i by Cardiologist; Test type: Other; p = 0.0401, Fisher Exact

31. Secondary Outcome: Number of Patients With Any Type of Cardiovascular Disease (CVD)
Description: Number of patients with cardiovascular disease (CVD) is reported. Patients with cardiovascular disease were considered patients for whom 'History of acute myocardial infarction', 'History of cardiology intervention', 'Ischemic heart disease', 'Congestive heart failure', 'History of stroke' or 'Peripheral arterial disease', were documented as comorbidities.
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | T2D Patients From Central Eastern Europe
Number analyzed (Participants) | 4055
Participants | 1485

32. Secondary Outcome: Number of Patients With Chronic Kidney Disease (CKD) by Physician's Assessment
Description: Number of patients with chronic kidney disease (CKD) by physician's assessment (patients for whom CKD was reported as a comorbidity) is reported.
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | T2D Patients From Central Eastern Europe
Number analyzed (Participants) | 4055
Participants | 586

33. Secondary Outcome: Number of Patients With Documentation of Estimated Glomerular Filtration Rate (eGFR) / Urine Albumin Creatinine Ratio (UACR) Status
Description: Number of patients with documentation of estimated Glomerular Filtration Rate (eGFR) / Urine Albumin Creatinine Ratio (UACR) status is reported.
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | T2D Patients From Central Eastern Europe
Number analyzed (Participants) | 4055
Participants | 3175

34. Secondary Outcome: Number of Patients With Chronic Kidney Disease (CKD) by Estimated Glomerular Filtration Rate (eGFR) and Urine Albumin Creatinine Ratio (UACR) Status
Description: Number of patients with Chronic Kidney Disease (CKD) by estimated Glomerular Filtration Rate (eGFR) and Urine Albumin Creatinine Ratio (UACR) status is reported.
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: Patients in the Prescribed patient set (PPS) (all patients fulfilling inclusion and exclusion criteria who have received a first prescription of a respective type 2 diabetes (T2D) medication and whose documentation was electronically signed by the physician) with documentation of of eGFR / UACR status.
Measure: Count of Participants; unit: Participants
Arm/Group | T2D Patients From Central Eastern Europe
Number analyzed (Participants) | 3175
Participants | 886

35. Secondary Outcome: Number of Patients in Each Category of the Different Types of Cardiovascular Disease
Description: Number of patients in each category of the different types of cardiovascular disease is reported.
  The following types of cardiovascular diseases are reported:
  * Myocardial infarction
  * Cardiology intervention (Percutaneous Coronary Intervention (PCI) or Coronary Artery Bypass Grafting (CABG))
  * Ischemic heart disease
  * Congestive heart failure
  * Stroke
  * Peripheral arterial disease
  The categories reported for each type of cardiovascular disease are:
  * Yes
  * No
  * Unknown
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | T2D Patients From Central Eastern Europe
Number analyzed (Participants) | 4055
Participants
  Myocardial infarction: Yes | 450
  Myocardial infarction: No | 3558
  Myocardial infarction: Unknown | 47
  Cardiology intervention (PCI or CABG): Yes | 525
  Cardiology intervention (PCI or CABG): No | 3471
  Cardiology intervention (PCI or CABG): Unknown | 59
  Ischemic heart disease: Yes | 1087
  Ischemic heart disease: No | 2910
  Ischemic heart disease: Unknown | 58
  Congestive heart failure: Yes | 421
  Congestive heart failure: No | 3511
  Congestive heart failure: Unknown | 123
  Stroke: Yes | 248
  Stroke: No | 3764
  Stroke: Unknown | 43
  Peripheral arterial disease: Yes | 350
  Peripheral arterial disease: No | 3643
  Peripheral arterial disease: Unknown | 62

36. Secondary Outcome: Number of Patients in Each Category of the Different Types of Congestive Heart Failure (CHF) - Confirmed by Echocardiography
Description: Number of patients in each category of the different types of congestive heart failure (CHF) which was confirmed by echocardiography is reported.
  The reported categories of congestive heart failure confirmed by echocardiography are:
  * Yes
  * No
  * Unknown
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: Patients in the Prescribed patient set (PPS) (all patients fulfilling inclusion and exclusion criteria who have received a first prescription of a respective type 2 diabetes (T2D) medication and whose documentation was electronically signed by the physician) with congestive heart failure.
Measure: Count of Participants; unit: Participants
Arm/Group | T2D Patients From Central Eastern Europe
Number analyzed (Participants) | 421
Participants
  Yes | 245
  No | 86
  Unknown | 90

37. Secondary Outcome: Number of Patients With Any Type of Cardiovascular Disease (CVD) and Without CVD According to Prescribing Specialist
Description: Number of patients with any type of cardiovascular disease (CVD) or without CVD according to prescribing specialist is reported. Patients with cardiovascular disease were considered patients for whom 'History of acute myocardial infarction', 'History of cardiology intervention', 'Ischemic heart disease', 'Congestive heart failure', 'History of stroke' or 'Peripheral arterial disease', were documented as comorbidities.
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on T2D Medication by Endocrinologist | Patients Initiated on T2D Medication by Diabetologist | Patients Initiated on T2D Medication by Cardiologist
Number analyzed (Participants) | 1652 | 2301 | 102
Participants
  Patients with any type of CVD | 736 | 656 | 93
  Patients without CVD | 916 | 1645 | 9

38. Secondary Outcome: Number of Patients With Chronic Kidney (CKD) (Patients for Whom CKD Was Reported as a Comorbidity) or Without CKD by Physician's Assessment According to Prescribing Specialist
Description: Number of patients with chronic kidney (CKD) and without CKD by physician's assessment according to prescribing specialist is reported.
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on T2D Medication by Endocrinologist | Patients Initiated on T2D Medication by Diabetologist | Patients Initiated on T2D Medication by Cardiologist
Number analyzed (Participants) | 1652 | 2301 | 102
Participants
  Patients with CKD by physician's assessment | 327 | 244 | 15
  Patients without CKD by physician's assessment | 1325 | 2057 | 87

39. Secondary Outcome: Number of Patients With Chronic Kidney Disease (CKD) by eGFR and UACR Status According to Prescribing Specialist
Description: Number of patients with chronic kidney disease (CKD) by estimated Glomerular Filtration Rate (eGFR) and Urine Albumin Creatinine Ratio (UACR) status - according to prescribing specialist is reported.
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: Patients in the Prescribed patient set (PPS) (all patients fulfilling inclusion and exclusion criteria who have received a first prescription of a respective type 2 diabetes (T2D) medication and whose documentation was electronically signed by the physician) with documentation of eGFR and/or UACR status are reported.
Measure: Count of Participants; unit: Participants
Groups:
- Patients Initiated on T2D Medication by Cardiologist: Patients with type 2 diabetes (T2D) from Central Eastern Europe (CEE) (Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who were newly initiated (first ever use) empagliflozin or other sodium dependent glucose transporter inhibitor (SGLT2i), dipeptidyl peptidase 4 inhibitor (DPP4i) or glucagon-like peptide-1 receptor agonist (GLP-1 RA) by cardiologist between September 2018 and December 2018 (study index date 1).
Arm/Group | Patients Initiated on T2D Medication by Endocrinologist | Patients Initiated on T2D Medication by Diabetologist | Patients Initiated on T2D Medication by Cardiologist
Number analyzed (Participants) | 1493 | 1604 | 78
Participants | 508 | 358 | 20

40. Secondary Outcome: Number of Patients With or Without at Least One Cardiovascular Disease (CVD) Type According to Type 2 Diabetes (T2D) Medication Initiated at Study Index Date 1
Description: Number of patients with or without at least one cardiovascular disease (CVD) type according to type 2 diabetes (T2D) medication initiated at study index date 1 is reported.
  Patients with cardiovascular disease were considered patients for whom 'History of acute myocardial infarction', 'History of cardiology intervention', 'Ischemic heart disease', 'Congestive heart failure', 'History of stroke' or 'Peripheral arterial disease', were documented as comorbidities.
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Patients Initiated on Empagliflozin: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on empagliflozin between September 2018 and December 2018 (study index date 1).
- Patients Initiated on DPP4i: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on dipeptidyl peptidase 4 inhibitor (DPP4i) between September 2018 and December 2018 (study index date 1).
- Patients Initiated on GLP-1 RA: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on glucagon-like peptide-1 receptor agonist (GLP-1 RA) between September 2018 and December 2018 (study index date 1).
- Patients Initiated on Other SGLT2i: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on other sodium dependent glucose transporter inhibitor (SGLT2i) between September 2018 and December 2018 (study index date 1).
Arm/Group | Patients Initiated on Empagliflozin | Patients Initiated on DPP4i | Patients Initiated on GLP-1 RA | Patients Initiated on Other SGLT2i
Number analyzed (Participants) | 1966 | 1144 | 361 | 584
Participants
  Yes | 812 | 398 | 75 | 200
  No | 1154 | 746 | 286 | 384

41. Secondary Outcome: Number of Patients in Each Category of Different Types of Cardiovascular Disease (CVD) According to Type 2 Diabetes (T2D) Medication Initiated at Study Index Date 1
Description: Number of patients in each category of different types of cardiovascular disease (CVD) according to type 2 diabetes (T2D) medication initiated at study index date 1 is reported.
  The following types of cardiovascular diseases are reported:
  * Myocardial infarction
  * Cardiology intervention (Percutaneous Coronary Intervention (PCI) or Coronary Artery Bypass Grafting (CABG))
  * Ischemic heart disease
  * Congestive heart failure
  * Stroke
  * Peripheral arterial disease
  The categories reported for each type of cardiovascular disease are:
  * Yes
  * No
  * Unknown
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on Empagliflozin | Patients Initiated on DPP4i | Patients Initiated on GLP-1 RA | Patients Initiated on Other SGLT2i
Number analyzed (Participants) | 1966 | 1144 | 361 | 584
Participants
  Myocardial infarction: Yes | 276 | 91 | 22 | 61
  Myocardial infarction: No | 1667 | 1039 | 334 | 518
  Myocardial infarction: Unknown | 23 | 14 | 5 | 5
  Cardiology intervention (PCI or CABG): Yes | 328 | 98 | 30 | 69
  Cardiology intervention (PCI or CABG): No | 1614 | 1024 | 324 | 509
  Cardiology intervention (PCI or CABG): Unknown | 24 | 22 | 7 | 6
  Ischemic heart disease: Yes | 631 | 265 | 50 | 141
  Ischemic heart disease: No | 1312 | 860 | 305 | 433
  Ischemic heart disease: Unknown | 23 | 19 | 6 | 10
  Congestive heart failure: Yes | 252 | 104 | 14 | 51
  Congestive heart failure: No | 1664 | 997 | 337 | 513
  Congestive heart failure: Unknown | 50 | 43 | 10 | 20
  Stroke: Yes | 128 | 76 | 12 | 32
  Stroke: No | 1819 | 1056 | 342 | 547
  Stroke: Unknown | 19 | 12 | 7 | 5
  Peripheral arterial disease: Yes | 171 | 118 | 15 | 46
  Peripheral arterial disease: No | 1767 | 1008 | 339 | 529
  Peripheral arterial disease: Unknown | 28 | 18 | 7 | 9

42. Secondary Outcome: Number of Patients in Each Category of Congestive Heart Failure (CHF) Confirmed by Echocardiography According to Type 2 Diabetes (T2D) Medication Initiated at Study Index Date 1
Description: Number of patients in each category of congestive heart failure (CHF) confirmed by echocardiography according to type 2 diabetes (T2D) medication initiated at study index date 1 is reported.
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for outcome 36
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on Empagliflozin | Patients Initiated on DPP4i | Patients Initiated on GLP-1 RA | Patients Initiated on Other SGLT2i
Number analyzed (Participants) | 252 | 104 | 14 | 51
Participants
  Yes | 164 | 42 | 9 | 30
  No | 36 | 39 | 4 | 7
  Unknown | 52 | 23 | 1 | 14

43. Secondary Outcome: Number of Patients With or Without at Least One Cardiovascular Disease (CVD) Type According to Type 2 Diabetes (T2D) Medication for the Patients Who Were Initiated on T2D Medication From by Endocrinologist
Description: Number of patients with or without at least one cardiovascular disease (CVD) type according to type 2 diabetes (T2D) medication for the patients who were initiated on T2D medication by endocrinologist is reported. Patients with cardiovascular disease were considered patients for whom 'History of acute myocardial infarction', 'History of cardiology intervention', 'Ischemic heart disease', 'Congestive heart failure', 'History of stroke' or 'Peripheral arterial disease', were documented as comorbidities.
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on Empagliflozin by Endocrinologist | Patients Initiated on DPP4i by Endocrinologist | Patients Initiated on GLP-1 RA by Endocrinologist | Patients Initiated on Other SGLT2i by Endocrinologist
Number analyzed (Participants) | 815 | 504 | 89 | 244
Participants
  Yes | 380 | 229 | 28 | 99
  No | 435 | 275 | 61 | 145

44. Secondary Outcome: Number of Patients With or Without at Least One Cardiovascular Disease (CVD) Type According to Type 2 Diabetes (T2D) Medication for the Patients Who Were Initiated on T2D Medication by Diabetologist
Description: Number of patients with or without at least one cardiovascular disease (CVD) type according to type 2 diabetes (T2D) medication for the patients who were initiated on T2D medication by diabetologist is reported. Patients with cardiovascular disease were considered patients for whom 'History of acute myocardial infarction', 'History of cardiology intervention', 'Ischemic heart disease', 'Congestive heart failure', 'History of stroke' or 'Peripheral arterial disease', were documented as comorbidities.
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Groups:
- Patients Initiated on Other SGLT2i by Diabetologist: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) with other sodium dependent glucose transporter inhibitor (SGLT2i) between September 2018 and December 2018 (study index date 1) by diabetologist.
Arm/Group | Patients Initiated on Empagliflozin by Diabetologist | Patients Initiated on DPP4i by Diabetologist | Patients Initiated on GLP-1 RA by Diabetologist | Patients Initiated on Other SGLT2i by Diabetologist
Number analyzed (Participants) | 1073 | 624 | 271 | 333
Participants
  Yes | 362 | 154 | 46 | 94
  No | 711 | 470 | 225 | 239

45. Secondary Outcome: Number of Patients With or Without at Least One Cardiovascular Disease (CVD) Type According to Type 2 Diabetes (T2D) Medication for the Patients Who Were Initiated on T2D Medication by Cardiologist
Description: Number of patients with or without at least one cardiovascular disease (CVD) type according to type 2 diabetes (T2D) medication for the patients who were initiated on T2D medication by cardiologist is reported. Patients with cardiovascular disease were considered patients for whom 'History of acute myocardial infarction', 'History of cardiology intervention', 'Ischemic heart disease', 'Congestive heart failure', 'History of stroke' or 'Peripheral arterial disease', were documented as comorbidities.
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on Empagliflozin by Cardiologist | Patients Initiated on DPP4i by Cardiologist | Patients Initiated on GLP-1 RA by Cardiologist | Patients Initiated on Other SGLT2i by Cardiologist
Number analyzed (Participants) | 78 | 16 | 1 | 7
Participants
  Yes | 70 | 15 | 1 | 7
  No | 8 | 1 | 0 | 0

46. Secondary Outcome: Number of Patients With Chronic Kidney (CKD) or Without CKD by Physician's Assessment According to Type 2 Diabetes (T2D) Medication Initiated at Study Index Date 1
Description: Number of patients with chronic kidney (CKD) (patients for whom CKD was reported as a comorbidity) or without CKD by physician's assessment according to type 2 diabetes (T2D) medication initiated at study index date 1 is reported.
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on Empagliflozin | Patients Initiated on DPP4i | Patients Initiated on GLP-1 RA | Patients Initiated on Other SGLT2i
Number analyzed (Participants) | 1966 | 1144 | 361 | 584
Participants
  Patients with CKD by physician's assessment | 221 | 289 | 26 | 50
  Patients without CKD by physician's assessment | 1745 | 855 | 335 | 534

47. Secondary Outcome: Number of Patients With Chronic Kidney (CKD) and Without CKD by eGFR and UACR Status According to Type 2 Diabetes (T2D) Medication Initiated at Study Index Date 1
Description: Number of patients with chronic kidney (CKD) (patients for whom CKD was reported as a comorbidity) and without CKD by estimated Glomerular Filtration Rate (eGFR) and Urine Albumin Creatinine Ratio (UACR) status according to type 2 diabetes (T2D) medication initiated at study index date 1 is reported.
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: Patients in the prescribed patient set (PPS) with available eGFR and UACR status. PPS included all patients fulfilling inclusion and exclusion criteria who have received a first prescription of a respective type 2 diabetes (T2D) medication and whose documentation was electronically signed by the physician.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on Empagliflozin | Patients Initiated on DPP4i | Patients Initiated on GLP-1 RA | Patients Initiated on Other SGLT2i
Number analyzed (Participants) | 1568 | 907 | 265 | 435
Participants
  Patients with CKD by eGFR and UACR status | 386 | 365 | 50 | 85
  Patients without CKD by eGFR and UACR status | 1182 | 542 | 215 | 350

48. Secondary Outcome: Number of Patients in Each Category of Employment Status According to Type 2 Diabetes (T2D) Medication Initiated at Study Index Date 1
Description: Number of patients in each category of employment status according to type 2 diabetes (T2D) medication initiated at study index date 1 is reported.
  The categories of employment status are:
  * Employed
  * Not employed
  * Unknown
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on Empagliflozin | Patients Initiated on DPP4i | Patients Initiated on GLP-1 RA | Patients Initiated on Other SGLT2i
Number analyzed (Participants) | 1966 | 1144 | 361 | 584
Participants
  Employed | 966 | 433 | 229 | 302
  Not employed | 878 | 639 | 111 | 261
  Unknown | 122 | 72 | 21 | 21
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin vs Patients Initiated on DPP4i vs Patients Initiated on GLP-1 RA vs Patients Initiated on Other SGLT2i; Test type: Other; p < .0001, Chi-squared

49. Secondary Outcome: Number of Patients in Each Category of Family Status According to Type 2 Diabetes (T2D) Medication Initiated at Study Index Date 1
Description: Number of patients in each category of family status according to type 2 diabetes (T2D) medication initiated at study index date 1 is reported.
  The categories of family status are:
  * Single
  * Married
  * Divorced
  * Widowed
  * Unknown
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on Empagliflozin | Patients Initiated on DPP4i | Patients Initiated on GLP-1 RA | Patients Initiated on Other SGLT2i
Number analyzed (Participants) | 1966 | 1144 | 361 | 584
Participants
  Single | 124 | 86 | 26 | 42
  Married | 1339 | 668 | 252 | 411
  Divorced | 88 | 59 | 27 | 37
  Widowed | 143 | 147 | 19 | 31
  Unknown | 272 | 184 | 37 | 63
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin vs Patients Initiated on DPP4i vs Patients Initiated on GLP-1 RA vs Patients Initiated on Other SGLT2i; Test type: Other; p < .0001, Chi-squared

50. Secondary Outcome: Number of Patients in Each Category of Insurance Status According to Type 2 Diabetes (T2D) Medication Initiated at Study Index Date 1
Description: Number of patients in each category of insurance status according to type 2 diabetes (T2D) medication initiated at study index date 1 is reported.
  The categories of insurance status are:
  * Not insured
  * Statutory insured
  * Privately insured
  * Unknown
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on Empagliflozin | Patients Initiated on DPP4i | Patients Initiated on GLP-1 RA | Patients Initiated on Other SGLT2i
Number analyzed (Participants) | 1966 | 1144 | 361 | 584
Participants
  Not insured | 50 | 13 | 3 | 11
  Statutory insured | 1725 | 1055 | 336 | 539
  Privately insured | 89 | 35 | 13 | 16
  Unknown | 102 | 41 | 9 | 18
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin vs Patients Initiated on DPP4i vs Patients Initiated on GLP-1 RA vs Patients Initiated on Other SGLT2i; Test type: Other; p = 0.0008, Chi-squared

51. Secondary Outcome: Number of Patients in Each Category of Employment Status According to Type 2 Diabetes (T2D) Medication for the Patients Who Were Initiated on T2D Medication by Endocrinologist
Description: Number of patients in each category of employment status according to type 2 diabetes (T2D) medication for the patients who were initiated on T2D medication by endocrinologist is reported.
  The categories of employment status are:
  * Employed
  * Not employed
  * Unknown
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on Empagliflozin by Endocrinologist | Patients Initiated on DPP4i by Endocrinologist | Patients Initiated on GLP-1 RA by Endocrinologist | Patients Initiated on Other SGLT2i by Endocrinologist
Number analyzed (Participants) | 815 | 504 | 89 | 244
Participants
  Employed | 438 | 199 | 69 | 128
  Not employed | 345 | 286 | 17 | 109
  Unknown | 32 | 19 | 3 | 7

52. Secondary Outcome: Number of Patients in Each Category of Family Status According to Type 2 Diabetes (T2D) Medication for the Patients Who Were Initiated on T2D Medication by Endocrinologist
Description: Number of patients in each category of family status according to type 2 diabetes (T2D) medication for the patients who were initiated on T2D medication by endocrinologist is reported.
  The categories of family status are:
  * Single
  * Married
  * Divorced
  * Widowed
  * Unknown
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on Empagliflozin by Endocrinologist | Patients Initiated on DPP4i by Endocrinologist | Patients Initiated on GLP-1 RA by Endocrinologist | Patients Initiated on Other SGLT2i by Endocrinologist
Number analyzed (Participants) | 815 | 504 | 89 | 244
Participants
  Single | 55 | 52 | 7 | 22
  Married | 566 | 290 | 68 | 175
  Divorced | 44 | 27 | 5 | 6
  Widowed | 67 | 69 | 2 | 9
  Unknown | 83 | 66 | 7 | 32
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Endocrinologist vs Patients Initiated on DPP4i by Endocrinologist vs Patients Initiated on GLP-1 RA by Endocrinologist vs Patients Initiated on Other SGLT2i by Endocrinologist; Test type: Other; p < .0001, Chi-squared

53. Secondary Outcome: Number of Patients in Each Category of Insurance Status According to Type 2 Diabetes (T2D) Medication for the Patients Who Were Initiated on T2D Medication by Endocrinologist
Description: Number of patients in each category of insurance status according to type 2 diabetes (T2D) medication for the patients who were initiated on T2D medication by endocrinologist is reported.
  The categories of insurance status are:
  * Not insured
  * Statutory insured
  * Privately insured
  * Unknown
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on Empagliflozin by Endocrinologist | Patients Initiated on DPP4i by Endocrinologist | Patients Initiated on GLP-1 RA by Endocrinologist | Patients Initiated on Other SGLT2i by Endocrinologist
Number analyzed (Participants) | 815 | 504 | 89 | 244
Participants
  Not insured | 40 | 12 | 3 | 11
  Statutory insured | 630 | 438 | 73 | 208
  Privately insured | 82 | 34 | 13 | 16
  Unknown | 63 | 20 | 0.0 | 9
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Endocrinologist vs Patients Initiated on DPP4i by Endocrinologist vs Patients Initiated on GLP-1 RA by Endocrinologist vs Patients Initiated on Other SGLT2i by Endocrinologist; Test type: Other; p = 0.0001, Chi-squared

54. Secondary Outcome: Number of Patients in Each Category of Employment Status According to Type 2 Diabetes (T2D) Medication for the Patients Who Were Initiated on T2D Medication by Diabetologist
Description: Number of patients in each category of employment status according to type 2 diabetes (T2D) medication for the patients who were initiated on T2D medication by diabetologist is reported.
  The categories of employment status are:
  * Employed
  * Not employed
  * Unknown
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on Empagliflozin by Diabetologist | Patients Initiated on DPP4i by Diabetologist | Patients Initiated on GLP-1 RA by Diabetologist | Patients Initiated on Other SGLT2i by Diabetologist
Number analyzed (Participants) | 1073 | 624 | 271 | 333
Participants
  Employed | 491 | 228 | 159 | 171
  Not employed | 500 | 345 | 94 | 150
  Unknown | 82 | 51 | 18 | 12
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Diabetologist vs Patients Initiated on DPP4i by Diabetologist vs Patients Initiated on GLP-1 RA by Diabetologist vs Patients Initiated on Other SGLT2i by Diabetologist; Test type: Other; p < .0001, Chi-squared

55. Secondary Outcome: Number of Patients in Each Category of Family Status According to Type 2 Diabetes (T2D) Medication for the Patients Who Were Initiated on T2D Medication by Diabetologist
Description: Number of patients in each category of family status according to type 2 diabetes (T2D) medication for the patients who were initiated on T2D medication by diabetologist is reported.
  The categories of family status are:
  * Single
  * Married
  * Divorced
  * Widowed
  * Unknown
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on Empagliflozin by Diabetologist | Patients Initiated on DPP4i by Diabetologist | Patients Initiated on GLP-1 RA by Diabetologist | Patients Initiated on Other SGLT2i by Diabetologist
Number analyzed (Participants) | 1073 | 624 | 271 | 333
Participants
  Single | 56 | 33 | 19 | 19
  Married | 727 | 368 | 183 | 233
  Divorced | 38 | 31 | 22 | 31
  Widowed | 71 | 76 | 17 | 21
  Unknown | 181 | 116 | 30 | 29
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Diabetologist vs Patients Initiated on DPP4i by Diabetologist vs Patients Initiated on GLP-1 RA by Diabetologist vs Patients Initiated on Other SGLT2i by Diabetologist; Test type: Other; p < .0001, Chi-squared

56. Secondary Outcome: Number of Patients in Each Category of Insurance Status According to Type 2 Diabetes (T2D) Medication for the Patients Who Were Initiated on T2D Medication by Diabetologist
Description: Number of patients in each category of insurance status according to type 2 diabetes (T2D) medication for the patients who were initiated on T2D medication by diabetologist is reported.
  The categories of insurance status are:
  * Not insured
  * Statutory insured
  * Privately insured
  * Unknown
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Groups:
- Patients Initiated on Empagliflozin by Diabetologist: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) with empagliflozin between September 2018 and December 2018 (study index date 1) from diabetologist.
Arm/Group | Patients Initiated on Empagliflozin by Diabetologist | Patients Initiated on DPP4i by Diabetologist | Patients Initiated on GLP-1 RA by Diabetologist | Patients Initiated on Other SGLT2i by Diabetologist
Number analyzed (Participants) | 1073 | 624 | 271 | 333
Participants
  Not insured | 2 | 1 | 0.0 | 0.0
  Statutory insured | 1039 | 603 | 262 | 326
  Privately insured | 3 | 1 | 0.0 | 0
  Unknown | 29 | 19 | 9 | 7
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Diabetologist vs Patients Initiated on DPP4i by Diabetologist vs Patients Initiated on GLP-1 RA by Diabetologist vs Patients Initiated on Other SGLT2i by Diabetologist; Test type: Other; p = 0.9184, Chi-squared
Statistical Analysis 2: Comparison: Patients Initiated on Empagliflozin by Diabetologist vs Patients Initiated on DPP4i by Diabetologist vs Patients Initiated on GLP-1 RA by Diabetologist vs Patients Initiated on Other SGLT2i by Diabetologist; Test type: Other; p = 0.9911, Fisher Exact

57. Secondary Outcome: Number of Patients in Each Category of Employment Status According to Type 2 Diabetes (T2D) Medication for the Patients Who Were Initiated on T2D Medication by Cardiologist
Description: Number of patients in each category of employment status according to type 2 diabetes (T2D) medication for the patients who were initiated on T2D medication by cardiologist is reported.
  The categories of employment status are:
  * Employed
  * Not employed
  * Unknown
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on Empagliflozin by Cardiologist | Patients Initiated on DPP4i by Cardiologist | Patients Initiated on GLP-1 RA by Cardiologist | Patients Initiated on Other SGLT2i by Cardiologist
Number analyzed (Participants) | 78 | 16 | 1 | 7
Participants
  Employed | 37 | 6 | 1 | 3
  Not employed | 33 | 8 | 0 | 2
  Unknown | 8 | 2 | 0 | 2
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Cardiologist vs Patients Initiated on DPP4i by Cardiologist vs Patients Initiated on GLP-1 RA by Cardiologist vs Patients Initiated on Other SGLT2i by Cardiologist; Test type: Other; p = 0.6967, Chi-squared
Statistical Analysis 2: Comparison: Patients Initiated on Empagliflozin by Cardiologist vs Patients Initiated on DPP4i by Cardiologist vs Patients Initiated on GLP-1 RA by Cardiologist vs Patients Initiated on Other SGLT2i by Cardiologist; Test type: Other; p = 0.6439, Fisher Exact

58. Secondary Outcome: Number of Patients in Each Category of Family Status According to Type 2 Diabetes (T2D) Medication for the Patients Who Were Initiated on T2D Medication by Cardiologist
Description: Number of patients in each category of family status according to type 2 diabetes (T2D) medication for the patients who were initiated on T2D medication by cardiologist is reported.
  The categories of family status are:
  * Single
  * Married
  * Divorced
  * Widowed
  * Unknown
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on Empagliflozin by Cardiologist | Patients Initiated on DPP4i by Cardiologist | Patients Initiated on GLP-1 RA by Cardiologist | Patients Initiated on Other SGLT2i by Cardiologist
Number analyzed (Participants) | 78 | 16 | 1 | 7
Participants
  Single | 13 | 1 | 0 | 1
  Married | 46 | 10 | 1 | 3
  Divorced | 6 | 1 | 0 | 0
  Widowed | 5 | 2 | 0 | 1
  Unknown | 8 | 2 | 0 | 2
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Cardiologist vs Patients Initiated on DPP4i by Cardiologist vs Patients Initiated on GLP-1 RA by Cardiologist vs Patients Initiated on Other SGLT2i by Cardiologist; Test type: Other; p = 0.9414, Chi-squared
Statistical Analysis 2: Comparison: Patients Initiated on Empagliflozin by Cardiologist vs Patients Initiated on DPP4i by Cardiologist vs Patients Initiated on GLP-1 RA by Cardiologist vs Patients Initiated on Other SGLT2i by Cardiologist; Test type: Other; p = 0.8142, Fisher Exact

59. Secondary Outcome: Number of Patients in Each Category of Insurance Status According to Type 2 Diabetes (T2D) Medication for the Patients Who Were Initiated on T2D Medication by Cardiologist
Description: Number of patients in each category of insurance status according to type 2 diabetes (T2D) medication for the patients who were initiated on T2D medication by cardiologist is reported.
  The categories of insurance status are:
  * Not insured
  * Statutory insured
  * Privately insured
  * Unknown
Time Frame: At study index date 1 (i.e. between September 2018 and December 2018).
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on Empagliflozin by Cardiologist | Patients Initiated on DPP4i by Cardiologist | Patients Initiated on GLP-1 RA by Cardiologist | Patients Initiated on Other SGLT2i by Cardiologist
Number analyzed (Participants) | 78 | 16 | 1 | 7
Participants
  Not insured | 8 | 0 | 0 | 0
  Statutory insured | 56 | 14 | 1 | 5
  Privately insured | 4 | 0 | 0 | 0
  Unknown | 10 | 2 | 0 | 2
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Cardiologist vs Patients Initiated on DPP4i by Cardiologist vs Patients Initiated on GLP-1 RA by Cardiologist vs Patients Initiated on Other SGLT2i by Cardiologist; Test type: Other; p = 0.7837, Chi-squared
Statistical Analysis 2: Comparison: Patients Initiated on Empagliflozin by Cardiologist vs Patients Initiated on DPP4i by Cardiologist vs Patients Initiated on GLP-1 RA by Cardiologist vs Patients Initiated on Other SGLT2i by Cardiologist; Test type: Other; p = 0.7538, Fisher Exact

60. Secondary Outcome: Number of Patients in Each Category of Status of Type 2 Diabetes (T2D) Medication at Index Date 2 According to Type 2 Diabetes (T2D) Medication Initiated at Study Index Date 1
Description: Number of patients in each category of status of type 2 diabetes (T2D) medication at index date 2 according to type 2 diabetes (T2D) medication initiated at study index date 1 is reported.
  The categories of status of T2D medication are:
  * Discontinued
  * Continued
Time Frame: At study index date 2 (= one year ± 2 months after index date 1 (study index date 1 was between September 2018 and December 2018)).
Population: Full Analysis set (FAS): All patients from Prescribed patient Set (PPS) with documentation at index date 2 and whose documentation was electronically signed by the physician. Patients included before the protocol amendment needed an additional signed informed consent at index date 2.
Measure: Count of Participants; unit: Participants
Groups:
- Patients Initiated on Empagliflozin: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on empagliflozin between September 2018 and December 2018 (study index date 1) and have consented to documentation at study index date 2.
- Patients Initiated on DPP4i: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on dipeptidyl peptidase 4 inhibitor (DPP4i) between September 2018 and December 2018 (study index date 1) and have consented to documentation at study index date 2.
- Patients Initiated on GLP-1 RA: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on glucagon-like peptide-1 receptor agonist (GLP-1 RA) between September 2018 and December 2018 (study index date 1) and have consented to documentation at study index date 2.
- Patients Initiated on Other SGLT2i: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on other sodium dependent glucose transporter inhibitor (SGLT2i) between September 2018 and December 2018 (study index date 1) and have consented to documentation at study index date 2.
Arm/Group | Patients Initiated on Empagliflozin | Patients Initiated on DPP4i | Patients Initiated on GLP-1 RA | Patients Initiated on Other SGLT2i
Number analyzed (Participants) | 1697 | 1053 | 332 | 536
Participants
  Discontinued | 134 | 129 | 38 | 60
  Continued | 1563 | 924 | 294 | 476
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin vs Patients Initiated on DPP4i vs Patients Initiated on GLP-1 RA vs Patients Initiated on Other SGLT2i; Test type: Other; p = 0.0012, Chi-squared

61. Secondary Outcome: Number of Patients in Each Category of Status of Type 2 Diabetes (T2D) Medication at Index Date 2 According to T2D Medication for the Patients Who Were Initiated on T2D Medication by Endocrinologist
Description: Number of patients in each category of status of type 2 diabetes (T2D) medication at index date 2 according to T2D medication for the patients who were initiated on T2D medication by endocrinologist is reported.
  The categories of status of T2D medication are:
  * Discontinued
  * Continued
Time Frame: as for outcome 60
Population: Patients of the full analysis set (FAS) who were initiated on type 2 diabetes (T2D) medication by endocrinologist. FAS included all patients from the prescribed patient set (PPS) with documentation at index date 2 and whose documentation was electronically signed by the physician. Patients included before the protocol amendment needed an additional signed informed consent at index date 2.
Measure: Count of Participants; unit: Participants
Groups:
- Patients Initiated on Empagliflozin by Endocrinologist: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on empagliflozin between September 2018 and December 2018 (study index date 1) by endocrinologist and have consented to documentation at study index date 2.
- Patients Initiated on DPP4i by Endocrinologist: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on dipeptidyl peptidase 4 inhibitor (DPP4i) between September 2018 and December 2018 (study index date 1) by endocrinologist and have consented to documentation at study index date 2.
- Patients Initiated on GLP-1 RA by Endocrinologist: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on glucagon-like peptide-1 receptor agonist (GLP-1 RA) between September 2018 and December 2018 (study index date 1) by endocrinologist and have consented to documentation at study index date 2.
- Patients Initiated on Other SGLT2i by Endocrinologist: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on other sodium dependent glucose transporter inhibitor (SGLT2i) between September 2018 and December 2018 (study index date 1) by endocrinologist and have consented to documentation at study index date 2.
Arm/Group | Patients Initiated on Empagliflozin by Endocrinologist | Patients Initiated on DPP4i by Endocrinologist | Patients Initiated on GLP-1 RA by Endocrinologist | Patients Initiated on Other SGLT2i by Endocrinologist
Number analyzed (Participants) | 731 | 479 | 81 | 214
Participants
  Discontinued | 42 | 58 | 17 | 26
  Continued | 689 | 421 | 64 | 188
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Endocrinologist vs Patients Initiated on DPP4i by Endocrinologist vs Patients Initiated on GLP-1 RA by Endocrinologist vs Patients Initiated on Other SGLT2i by Endocrinologist; Test type: Other; p < .0001, Chi-squared

62. Secondary Outcome: Number of Patients in Each Category of Status of Type 2 Diabetes (T2D) Medication at Index Date 2 According to T2D Medication for the Patients Who Were Initiated on T2D Medication by Diabetologist
Description: Number of patients in each category of status of type 2 diabetes (T2D) medication at index date 2 according to T2D medication for the patients who were initiated on T2D medication by diabetologist is reported.
  The categories of status of T2D medication are:
  * Discontinued
  * Continued
Time Frame: as for outcome 60
Population: Patients of the full analysis set (FAS) who were initiated on type 2 diabetes (T2D) medication by diabetologist. FAS included all patients from the prescribed patient set (PPS) with documentation at index date 2 and whose documentation was electronically signed by the physician. Patients included before the protocol amendment needed an additional signed informed consent at index date 2.
Measure: Count of Participants; unit: Participants
Groups:
- Patients Initiated on Empagliflozin by Diabetologist: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on empagliflozin between September 2018 and December 2018 (study index date 1) by diabetologist and have consented to documentation at study index date 2.
- Patients Initiated on DPP4i by Diabetologist: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on dipeptidyl peptidase 4 inhibitor (DPP4i) between September 2018 and December 2018 (study index date 1) by diabetologist and have consented to documentation at study index date 2.
- Patients Initiated on GLP-1 RA by Diabetologist: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) with glucagon-like peptide-1 receptor agonist (GLP-1 RA) between September 2018 and December 2018 (study index date 1) from diabetologist and have consented to documentation at study index date 2.
- Patients Initiated on Other SGLT2i by Diabetologist: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on other sodium dependent glucose transporter inhibitor (SGLT2i) between September 2018 and December 2018 (study index date 1) from diabetologist and have consented to documentation at study index date 2.
Arm/Group | Patients Initiated on Empagliflozin by Diabetologist | Patients Initiated on DPP4i by Diabetologist | Patients Initiated on GLP-1 RA by Diabetologist | Patients Initiated on Other SGLT2i by Diabetologist
Number analyzed (Participants) | 906 | 561 | 250 | 316
Participants
  Discontinued | 87 | 71 | 21 | 34
  Continued | 819 | 490 | 229 | 282
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Diabetologist vs Patients Initiated on DPP4i by Diabetologist vs Patients Initiated on GLP-1 RA by Diabetologist vs Patients Initiated on Other SGLT2i by Diabetologist; Test type: Other; p = 0.1906, Chi-squared

63. Secondary Outcome: Number of Patients in Each Category of Status of Type 2 Diabetes (T2D) Medication at Index Date 2 According to T2D Medication for the Patients Who Were Initiated on T2D Medication by Cardiologist
Description: Number of patients in each category of status of type 2 diabetes (T2D) medication at index date 2 according to T2D medication for the patients who were initiated on T2D medication by cardiologist is reported.
  The categories of status of T2D medication are:
  * Discontinued
  * Continued
Time Frame: as for outcome 60
Population: Patients of the full analysis set (FAS) who were initiated on type 2 diabetes (T2D) medication by cardiologist. FAS included all patients from the prescribed patient set (PPS) with documentation at index date 2 and whose documentation was electronically signed by the physician. Patients included before the protocol amendment needed an additional signed informed consent at index date 2.
Measure: Count of Participants; unit: Participants
Groups:
- Patients Initiated on Empagliflozin by Cardiologist: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on empagliflozin between September 2018 and December 2018 (study index date 1) by cardiologist and have consented to documentation at study index date 2.
- Patients Initiated on DPP4i by Cardiologist: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on dipeptidyl peptidase 4 inhibitor (DPP4i) between September 2018 and December 2018 (study index date 1) by cardiologist and have consented to documentation at study index date 2.
- Patients Initiated on GLP-1 RA by Cardiologist: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on glucagon-like peptide-1 receptor agonist (GLP-1 RA) between September 2018 and December 2018 (study index date 1) by cardiologist and have consented to documentation at study index date 2.
- Patients Initiated on Other SGLT2i by Cardiologist: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on other sodium dependent glucose transporter inhibitor (SGLT2i) between September 2018 and December 2018 (study index date 1) by cardiologist and have consented to documentation at study index date 2.
Arm/Group | Patients Initiated on Empagliflozin by Cardiologist | Patients Initiated on DPP4i by Cardiologist | Patients Initiated on GLP-1 RA by Cardiologist | Patients Initiated on Other SGLT2i by Cardiologist
Number analyzed (Participants) | 60 | 13 | 1 | 6
Participants
  Discontinued | 5 | 0 | 0 | 0
  Continued | 55 | 13 | 1 | 6
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Cardiologist vs Patients Initiated on DPP4i by Cardiologist vs Patients Initiated on GLP-1 RA by Cardiologist vs Patients Initiated on Other SGLT2i by Cardiologist; Test type: Other; p = 0.6198, Chi-squared
Statistical Analysis 2: Comparison: Patients Initiated on Empagliflozin by Cardiologist vs Patients Initiated on DPP4i by Cardiologist vs Patients Initiated on GLP-1 RA by Cardiologist vs Patients Initiated on Other SGLT2i by Cardiologist; Test type: Other; p = 0.7297, Fisher Exact

64. Secondary Outcome: Number of Patients in Each Category of Reason for Discontinuation of Type 2 Diabetes (T2D) Medication by Country
Description: Number of patients in each category of reason for discontinuation of type 2 diabetes (T2D) medication by country is reported.
  The categories of reason for discontinuation of T2D medication are:
  * Lack of efficacy
  * Medication administration
  * Financial burden regarding co-payment
  * Lost to follow-up
  * Adverse event
  * Other
Time Frame: as for outcome 60
Population: Patients in the full analysis set (FAS) who discontinued the study medication. FAS included all patients from the prescribed patient set (PPS) with documentation at index date 2 and whose documentation was electronically signed by the physician. Patients included before the protocol amendment needed an additional signed informed consent at index date 2.
Measure: Count of Participants; unit: Participants
Groups:
- T2D Patients From Bulgaria: Patients with type 2 diabetes (T2D) from Bulgaria who were newly initiated (first ever use) on empagliflozin or other sodium dependent glucose transporter inhibitor (SGLT2i), dipeptidyl peptidase 4 inhibitor (DPP4i) or glucagon-like peptide-1 receptor agonist (GLP-1 RA) between September 2018 and December 2018 (study index date 1) and have consented to documentation at study index date 2.
- T2D Patients From Czech Republic: Patients with type 2 diabetes (T2D) from Czech Republic who were newly initiated (first ever use) on empagliflozin or other sodium dependent glucose transporter inhibitor (SGLT2i), dipeptidyl peptidase 4 inhibitor (DPP4i) or glucagon-like peptide-1 receptor agonist (GLP-1 RA) between September 2018 and December 2018 (study index date 1) and have consented to documentation at study index date 2.
- T2D Patients From Hungary: Patients with type 2 diabetes (T2D) from Hungary who were newly initiated (first ever use) on empagliflozin or other sodium dependent glucose transporter inhibitor (SGLT2i), dipeptidyl peptidase 4 inhibitor (DPP4i) or glucagon-like peptide-1 receptor agonist (GLP-1 RA) between September 2018 and December 2018 (study index date 1) and have consented to documentation at study index date 2.
- T2D Patients From Poland: Patients with type 2 diabetes (T2D) from Poland who were newly initiated (first ever use) on empagliflozin or other sodium dependent glucose transporter inhibitor (SGLT2i), dipeptidyl peptidase 4 inhibitor (DPP4i) or glucagon-like peptide-1 receptor agonist (GLP-1 RA) between September 2018 and December 2018 (study index date 1) and have consented to documentation at study index date 2.
- T2D Patients From Russian Federation: Patients with type 2 diabetes (T2D) from Russian Federation who were newly initiated (first ever use) on empagliflozin or other sodium dependent glucose transporter inhibitor (SGLT2i), dipeptidyl peptidase 4 inhibitor (DPP4i) or glucagon-like peptide-1 receptor agonist (GLP-1 RA) between September 2018 and December 2018 (study index date 1) and have consented to documentation at study index date 2.
Arm/Group | T2D Patients From Bulgaria | T2D Patients From Czech Republic | T2D Patients From Hungary | T2D Patients From Poland | T2D Patients From Russian Federation
Number analyzed (Participants) | 25 | 90 | 16 | 104 | 126
Participants
  Lack of efficacy | 17 | 64 | 9 | 15 | 30
  Medication administration | 1 | 1 | 0 | 1 | 16
  Financial burden regarding co-payment | 2 | 0 | 2 | 58 | 60
  Lost to follow-up | 0 | 3 | 1 | 5 | 1
  Adverse event | 3 | 9 | 1 | 23 | 7
  Other | 2 | 13 | 3 | 2 | 12

65. Secondary Outcome: Number of Patients in Each Category of Reason for Discontinuation of Type 2 Diabetes (T2D) Medication According to Type 2 Diabetes (T2D) Medication Initiated at Study Index Date 1
Description: Number of patients in each category of reason for discontinuation of type 2 diabetes (T2D) medication according to type 2 diabetes (T2D) medication initiated at study index date 1 is reported.
  The categories of reason for discontinuation of T2D medication are:
  * Lack of efficacy
  * Medication administration
  * Financial burden regarding co-payment
  * Lost to follow-up
  * Adverse event
  * Other
Time Frame: as for outcome 60
Population: as for outcome 64
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on Empagliflozin | Patients Initiated on DPP4i | Patients Initiated on GLP-1 RA | Patients Initiated on Other SGLT2i
Number analyzed (Participants) | 134 | 129 | 38 | 60
Participants
  Lack of efficacy | 29 | 67 | 20 | 19
  Medication administration | 8 | 7 | 1 | 3
  Financial burden regarding co-payment | 49 | 37 | 9 | 27
  Lost to follow-up | 5 | 3 | 0 | 2
  Adverse event | 32 | 0 | 3 | 8
  Other | 11 | 15 | 5 | 1
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin vs Patients Initiated on DPP4i vs Patients Initiated on GLP-1 RA vs Patients Initiated on Other SGLT2i; Test type: Other; p < .0001, Chi-squared

66. Secondary Outcome: Number of Patients in Each Category of Reason for Discontinuation of Type 2 Diabetes (T2D) According to T2D Medication for the Patients Who Were Initiated on T2D Medication by Endocrinologist
Description: Number of patients in each category of reason for discontinuation of type 2 diabetes (T2D) according to T2D medication for the patients who were initiated on T2D medication by endocrinologist is reported.
  The categories of reason for discontinuation of T2D medication are:
  * Lack of efficacy
  * Medication administration
  * Financial burden regarding co-payment
  * Lost to follow-up
  * Adverse event
  * Other
Time Frame: as for outcome 60
Population: Patients in the full analysis set (FAS) who discontinued the study medication and who were initiated on type 2 diabetes (T2D) medication by endocrinologist. FAS included all patients from the prescribed patient set (PPS) with documentation at index date 2 and whose documentation was electronically signed by the physician. Patients included before the protocol amendment needed an additional signed informed consent at index date 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on Empagliflozin by Endocrinologist | Patients Initiated on DPP4i by Endocrinologist | Patients Initiated on GLP-1 RA by Endocrinologist | Patients Initiated on Other SGLT2i by Endocrinologist
Number analyzed (Participants) | 42 | 58 | 17 | 26
Participants
  Lack of efficacy | 10 | 26 | 6 | 2
  Medication administration | 6 | 6 | 0 | 3
  Financial burden regarding co-payment | 15 | 24 | 7 | 14
  Lost to follow-up | 1 | 0 | 0 | 0
  Adverse event | 2 | 0 | 2 | 6
  Other | 8 | 2 | 2 | 1
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Endocrinologist vs Patients Initiated on DPP4i by Endocrinologist vs Patients Initiated on GLP-1 RA by Endocrinologist vs Patients Initiated on Other SGLT2i by Endocrinologist; Test type: Other; p = 0.0012, Chi-squared
Statistical Analysis 2: Comparison: Patients Initiated on Empagliflozin by Endocrinologist vs Patients Initiated on DPP4i by Endocrinologist vs Patients Initiated on GLP-1 RA by Endocrinologist vs Patients Initiated on Other SGLT2i by Endocrinologist; Test type: Other; p = 0.0002, Fisher Exact

67. Secondary Outcome: Number of Patients in Each Category of Reason for Discontinuation of Type 2 Diabetes (T2D) Medication According to T2D Medication for the Patients Who Were Initiated on T2D Medication by Diabetologist
Description: Number of patients in each category of reason for discontinuation of type 2 diabetes (T2D) medication according to T2D medication for the patients who were initiated on T2D medication by diabetologist is reported.
  The categories of reason for discontinuation of T2D medication are:
  * Lack of efficacy
  * Medication administration
  * Financial burden regarding co-payment
  * Lost to follow-up
  * Adverse event
  * Other
Time Frame: as for outcome 60
Population: Patients in the full analysis set (FAS) who discontinued the study medication and who were initiated on type 2 diabetes (T2D) medication by diabetologist. FAS included all patients from the prescribed patient set (PPS) with documentation at index date 2 and whose documentation was electronically signed by the physician. Patients included before the protocol amendment needed an additional signed informed consent at index date 2.
Measure: Count of Participants; unit: Participants
Groups:
- Patients Initiated on GLP-1 RA by Diabetologist: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on glucagon-like peptide-1 receptor agonist (GLP-1 RA) between September 2018 and December 2018 (study index date 1) by diabetologist and have consented to documentation at study index date 2.
- Patients Initiated on Other SGLT2i by Diabetologist: Patients with type 2 diabetes from Central Eastern Europe (CEE) (i.e. Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who have been newly initiated (first ever use) on other sodium dependent glucose transporter inhibitor (SGLT2i) between September 2018 and December 2018 (study index date 1) by diabetologist and have consented to documentation at study index date 2.
Arm/Group | Patients Initiated on Empagliflozin by Diabetologist | Patients Initiated on DPP4i by Diabetologist | Patients Initiated on GLP-1 RA by Diabetologist | Patients Initiated on Other SGLT2i by Diabetologist
Number analyzed (Participants) | 87 | 71 | 21 | 34
Participants
  Lack of efficacy | 17 | 41 | 14 | 17
  Medication administration | 0 | 1 | 1 | 0
  Financial burden regarding co-payment | 34 | 13 | 2 | 13
  Lost to follow-up | 4 | 3 | 0 | 2
  Adverse event | 30 | 0 | 1 | 2
  Other | 2 | 13 | 3 | 0
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin by Diabetologist vs Patients Initiated on DPP4i by Diabetologist vs Patients Initiated on GLP-1 RA by Diabetologist vs Patients Initiated on Other SGLT2i by Diabetologist; Test type: Other; p < .0001, Chi-squared

68. Secondary Outcome: Number of Patients in Each Category of Reason for Discontinuation of Type 2 Diabetes (T2D) Medication According to T2D Medication for the Patients Who Were Initiated on T2D Medication by Cardiologist
Description: Number of patients in each category of reason for discontinuation of type 2 diabetes (T2D) medication according to T2D medication for the patients who were initiated on T2D medication by cardiologist is reported.
  The categories of reason for discontinuation of T2D medication are:
  * Lack of efficacy
  * Medication administration
  * Financial burden regarding co-payment
  * Lost to follow-up
  * Adverse event
  * Other
Time Frame: as for outcome 60
Population: Patients in the full analysis set (FAS) who discontinued the study medication and who were initiated on type 2 diabetes (T2D) medication by cardiologist. FAS included all patients from the prescribed patient set (PPS) with documentation at index date 2 and whose documentation was electronically signed by the physician. Patients included before the protocol amendment needed an additional signed informed consent at index date 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Initiated on Empagliflozin by Cardiologist | Patients Initiated on DPP4i by Cardiologist | Patients Initiated on GLP-1 RA by Cardiologist | Patients Initiated on Other SGLT2i by Cardiologist
Number analyzed (Participants) | 5 | 0 | 0 | 0
Participants
  Lack of efficacy | 2 |  |  |
  Medication administration | 2 |  |  |
  Financial burden regarding co-payment | 0 |  |  |
  Lost to follow-up | 0 |  |  |
  Adverse event | 0 |  |  |
  Other | 1 |  |  |

69. Secondary Outcome: Number of Patients for Each Type of Physician Specialties Involved in Decision for T2D Therapy Discontinuation According to Prescribing Specialist
Description: Number of patients for each type of physician specialties involved in decision for T2D therapy discontinuation according to prescribing specialist is reported.
Time Frame: as for outcome 60
Population: as for outcome 64
Measure: Count of Participants; unit: Participants
Groups:
- Patients Initiated on T2D Medication by Endocrinologist: Patients with type 2 diabetes (T2D) from Central Eastern Europe (CEE) (Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who were newly initiated (first ever use) on empagliflozin or other sodium dependent glucose transporter inhibitor (SGLT2i), dipeptidyl peptidase 4 inhibitor (DPP4i) or glucagon-like peptide-1 receptor agonist (GLP-1 RA) by endocrinologist between September 2018 and December 2018 (study index date 1) and have consented to documentation at study index date 2.
- Patients Initiated on T2D Medication by Diabetologist: Patients with type 2 diabetes (T2D) from Central Eastern Europe (CEE) (Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who were newly initiated (first ever use) on empagliflozin or other sodium dependent glucose transporter inhibitor (SGLT2i), dipeptidyl peptidase 4 inhibitor (DPP4i) or glucagon-like peptide-1 receptor agonist (GLP-1 RA) by diabetologist between September 2018 and December 2018 (study index date 1) and have consented to documentation at study index date 2.
- Patients Initiated on T2D Medication by Cardiologist: Patients with type 2 diabetes (T2D) from Central Eastern Europe (CEE) (Bulgaria, Czech Republic, Hungary, Poland and the Russian Federation) who were newly initiated (first ever use) on empagliflozin or other sodium dependent glucose transporter inhibitor (SGLT2i), dipeptidyl peptidase 4 inhibitor (DPP4i) or glucagon-like peptide-1 receptor agonist (GLP-1 RA) by cardiologist between September 2018 and December 2018 (study index date 1) and have consented to documentation at study index date 2.
Arm/Group | Patients Initiated on T2D Medication by Endocrinologist | Patients Initiated on T2D Medication by Diabetologist | Patients Initiated on T2D Medication by Cardiologist
Number analyzed (Participants) | 143 | 213 | 5
Participants
  Endocrinologist | 26 | 0 | 4
  Diabetologist | 0 | 2 | 0
  Cardiologist | 2 | 0 | 0
  General practitioner | 14 | 23 | 1
  Other | 2 | 3 | 0
  None | 102 | 185 | 0

70. Secondary Outcome: Time to Discontinuation of Type 2 Diabetes (T2D) Treatment According to Study Medication
Description: Time to discontinuation of type 2 diabetes (T2D) treatment according to study medication is reported.
  Time to discontinuation of T2D medication was estimated by Kaplan-Meier analysis. Patients who did not discontinue study medication at study index date 2 were censored.
Time Frame: From date of first prescription (study index date 1) to stop date of initial type 2 diabetes (T2D)) medication (documented at index date 2), up to 14 months..
Population: as for outcome 60
Measure: Mean (Standard Error); unit: months
Arm/Group | Patients Initiated on Empagliflozin | Patients Initiated on DPP4i | Patients Initiated on GLP-1 RA | Patients Initiated on Other SGLT2i
Number analyzed (Participants) | 1697 | 1053 | 332 | 536
months | 19.46 (0.73) | 18.28 (0.44) | 20.61 (0.62) | 14.04 (0.12)
Statistical Analysis 1: Comparison: Patients Initiated on Empagliflozin vs Patients Initiated on DPP4i vs Patients Initiated on GLP-1 RA vs Patients Initiated on Other SGLT2i; Test type: Other; p = 0.0030, Log Rank

ADVERSE EVENTS:
Time Frame: up to 14 months.
Description: Prescribed patient set (PPS): All patients fulfilling inclusion and exclusion criteria who have received a first prescription of a respective T2D medication and whose documentation was electronically signed by the physician.
  Within this observational study the seriousness of Adverse Events was not collected, therefore the "Total # at Risk by any Other Adverse Events" is "0". All adverse events collected in this study are reported under "Serious Adverse Events".
Arm/Group | T2D Patients From Central Eastern Europe
All-Cause Mortality (participants affected / at risk) | 0/4055
Serious Adverse Events (participants affected / at risk) | 43/4055
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | T2D Patients From Central Eastern Europe (N=4055)
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Thirst (General disorders) | 1
Genital infection (Infections and infestations) | 7
Infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 5
Vulvovaginal candidiasis (Infections and infestations) | 1
Vulvovaginitis (Infections and infestations) | 5
Glomerular filtration rate decreased (Investigations) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Dysuria (Renal and urinary disorders) | 11
Pollakiuria (Renal and urinary disorders) | 4
Balanoposthitis (Reproductive system and breast disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/40/NCT03807440/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/40/NCT03807440/SAP_001.pdf